CLINICAL TRIAL: NCT02446743
Title: A Phase 3b, Open Label, Controlled, Multi-Center, Extension Study to Assess the Persistence of Bactericidal Activity at 4 to 7.5 Years After Two Dose Primary Series of GlaxoSmithKline Biologicals Meningococcal B Recombinant Vaccine and the Response to a Third Dose in Adolescents and Young Adult Subjects Who Previously Participated in Parent Studies V72_41 (NCT01423084) and V72P10 (NCT00661713), Compared to Naïve Healthy Controls
Brief Title: Combined Study - Phase 3b MenB Long Term Persistence in Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 205218; V72_75 (Other: Novartis); 2017-000093-11 (EudraCT Number)
Record Dates: First submitted 2015-05-06; First posted 2015-05-18 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-04

CONDITIONS: Infections, Meningococcal
Keywords: Nervous System Diseases; Meningitis; Central Nervous System Diseases
MeSH Terms: conditions — Meningococcal Infections; Nervous System Diseases; Meningitis; Central Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 3B (Experimental): Subjects who received a third dose booster of rMenB+OMV NZ at 4 to 7.5 years after the last dose received during studies V72P10 (NCT00661713) or V72_41(NCT0142384), and had blood collected at baseline and at 3, 7 and 30 days after the third dose booster.
  Interventions: Biological: rMenB+OMV NZ (Meningococcal (Group B) multi component recombinant adsorbed vaccine)
- Group B_0_1 (Active Comparator): Subjects who received two doses of rMenB+OMV NZ at a 0 and 1 month schedule and had blood collected at baseline, 30 days after the first dose and 3 or 7, and 30 days after the second dose.
  Interventions: Biological: rMenB+OMV NZ (Meningococcal (Group B) multi component recombinant adsorbed vaccine)

INTERVENTIONS:
Biological: rMenB+OMV NZ (Meningococcal (Group B) multi component recombinant adsorbed vaccine) — One dose of the vaccine administered intramuscularly in the deltoid area of the non-dominant arm.

SUMMARY:
The purpose/aim of this study is to assess 1) the long-term persistence (4 to 7.5 years after the last dose) of bactericidal activity following primary vaccination with rMenB+OMV NZ in adolescents [who previously participated in parent studies V72_41 (NCT0142384) and V72P10 (NCT00661713)] and 2) the kinetics of immune response following booster vaccination with rMenB+OMV NZ

DETAILED DESCRIPTION:
After all subjects (Groups A and B) from Canada and Australia have completed the study, an interim analysis for the primary and secondary immunogenicity objectives will be performed. Follow on subjects (Group A) from parent study V72_41 (NCT0142384) will be analyzed for i) antibody persistence at approximately 4 years following a 2 dose primary series and ii) the immune response at 3, 7 and 30 days after a third dose (booster) of rMenB+OMV NZ. Canadian and Australian vaccine naïve subjects (Group B) will be analyzed for the immune response at 30 days after the first dose, and 3, 7 and 30 days after the second dose of rMenB+OMV NZ.

Subjects in Group B (naïve subjects) will be randomized into two different blood draw schedules according to a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criterion for follow-on subjects:
* Individuals who participated to Study V72_41 or V72P10 and have completed vaccination with rMenB+OMV NZ according to a 2-dose schedule

Inclusion Criterion for naïve subjects:

* Individuals of 15 through 21 years of age on the day of informed consent and assent as applicable (according to the subject's age) for subjects enrolled at sites that participated to Study V72_41.
* 17 through 24 years of age on the day of informed consent and assent as applicable (according to the subject's age) for subjects enrolled at sites that participated to Study V72P10.

Inclusion Criteria for all subjects:

* Individuals who have voluntarily given written informed consent after the nature of the study has been explained according to local regulatory requirements, prior to study entry.
* Individuals who can comply with study procedures including follow-up.
* Males Or Females of non-childbearing potential Or Females of childbearing potential who are using an effective birth control method .

Exclusion Criteria for all subjects

Exclusion Criterion for follow-on subjects:

• Received a third dose of a Meningococcal group B vaccine prior to enrolment in this study.

Exclusion Criterion for naïve subjects:

• Received any other Meningococcal group B vaccines prior to enrolment in this study.

Exclusion Criteria for all subjects:

* Progressive, unstable or uncontrolled clinical conditions.
* Hypersensitivity, including allergy, to any component of vaccines or medical equipment whose use is foreseen in this study.
* Abnormal function of the immune system.
* Received immunoglobulins or any blood products within 180 days prior to informed consent and assent as applicable (according to the subject's age).
* Received an investigational or non-registered medicinal product within 30 days prior to informed consent and assent as applicable (according to the subject's age).
* Study personnel as an immediate family or household member.
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the subject due to participation in the study.
* Positive results at the urine pregnancy test performed before study vaccination.

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 531 (Actual)
Dates: Start 2015-11-17 (Actual); Primary Completion 2016-09-23 (Actual); Study Completion 2016-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- Australia (4):
  - GSK Investigational Site, Sherwood, Queensland
  - GSK Investigational Site, North Adelaide, South Australia
  - GSK Investigational Site, Carlton, Victoria
  - GSK Investigational Site, Subiaco, Western Australia
- Canada (5):
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Newmarket, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Woodstock, Ontario
- GSK Investigational Site, Santiago, Chile

REFERENCES:
- [Derived] Nolan T, Santolaya ME, de Looze F, Marshall H, Richmond P, Henein S, Rheault P, Heaton K, Perrett KP, Garfield H, Gupta A, Ferguson M, D'Agostino D, Toneatto D, O'Ryan M. Antibody persistence and booster response in adolescents and young adults 4 and 7.5 years after immunization with 4CMenB vaccine. Vaccine. 2019 Feb 21;37(9):1209-1218. doi: 10.1016/j.vaccine.2018.12.059. Epub 2019 Jan 26. PMID 30691980

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 4 sites in Australia,6 sites in Canada & 2 sites in Chile.Analysis were performed on the study population (Groups 3B and B_0_1), but also repeated & stratified by parent study (i.e., V72_41 subjects using naïve subjects in Australia and Canada as controls, and V72P10 subjects using naïve subjects in Chile as controls)
Pre-assignment Details: All enrolled subjects were included in the study. Only groups 3B & B_0_1 were accounted for enrollment number as subjects from parent studies are included in the group 3B.
Groups:
- Group 3B: Subjects who received two doses of rMenB+OMV NZ administered at 0, 1 or 0,2 or 0,6 month schedule in study V72P10 and at 0,1 month schedule in study V72_41, and who received a third dose booster of rMenB+OMV NZ at 4 to 7.5 years after the last dose received during parent studies, and had blood collected at baseline and at 3, 7 and 30 days after the third dose booster.
- Group B_0_1: Naive subjects from Australia,Canada and Chile, who received two doses of rMenB+OMV NZ at a 0 and 1 month schedule and had blood collected at baseline, 30 days after the first dose and 3 or 7, and 30 days after the second dose.
Period: Overall Study
Arm/Group | Group 3B | Group B_0_1
Started | 276 | 255
Completed | 271 | 250
Not Completed | 5 | 5
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 1 | 1
Not completed — Other | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 3B | Group B_0_1 | Total
Number analyzed (Participants) | 276 | 255 | 531
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.5 (2.42) | 20.0 (2.69) | 19.7 (2.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 133 | 128 | 261
  Male | 143 | 127 | 270
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethinicity: American Indian or Alaska Native | 11 | 1 | 12
  Race/Ethinicity: Asian | 22 | 18 | 40
  Race/Ethinicity: Black or African American | 3 | 2 | 5
  Race/Ethinicity: Native Hawaiian or other Pacific Islander | 3 | 8 | 11
  Race/Ethinicity: White | 98 | 74 | 172
  Race/Ethinicity: Other | 139 | 152 | 291

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Human Serum Bactericidal Activity (hSBA)≥1:4
Description: Bactericidal activity was measured against the N. meningitidis group B indicator strains 5/99 and NZ98/254. This outcome measure was assessed only for strains 5/99 and NZ98/254.
Time Frame: Group 3B: Day 1 (prior to booster dose); Group B_0_1: Day 1 (prior to first dose).
Population: Analysis was performed on the Full analysis set (FAS) persistence. The FAS included all follow-on subjects (Group 3B) in the All Enrolled Set,& all naïve subjects (group B_0_1) in the All Enrolled Set who provided evaluable immunogenicity result at day 1,for at least one indicator strain.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Groups:
- Group 3B (V72_41): Subjects who received two doses of rMenB+OMV NZ administered at 0,1-month schedule in study V72_41 (NCT0142384) and who received a third dose booster of rMenB+OMV NZ at 4 to 7.5 years after the last dose received during study V72_41, and had blood collected at baseline and at 3, 7 and 30 days after the third dose booster.
- Group 3B (V72P10): Subjects who received two doses of rMenB+OMV NZ administered at 0,1 or 0,2 or 0,6 month schedule in study V72P10 (NCT00661713) and who received a third dose booster of rMenB+OMV NZ at 4 to 7.5 years after the last dose received during study V72P10, and had blood collected at baseline and at 3, 7 and 30 days after the third dose booster.
- Group 3B: Subjects who received two doses of rMenB+OMV NZ administered at 0, 1 or 0,2 or 0,6 month schedule in study V72P10 (NCT00661713) and at 0,1 month schedule in study V72_41(NCT0142384), and who received a third dose booster of rMenB+OMV NZ at 4 to 7.5 years after the last dose received during parent studies, and had blood collected at baseline and at 3, 7 and 30 days after the third dose booster.
- Group B_0_1 (V72_41): Naive subjects from Australia and Canada, who received two doses of rMenB+OMV NZ at a 0 and 1 month schedule in this study and had blood collected at baseline, 30 days after the first dose and 3 or 7, and 30 days after the second dose.
- Group B_0_1 (V72P10): Naive subjects from Chile, who received two doses of rMenB+OMV NZ at a 0 and 1 month schedule in this study and had blood collected at baseline, 30 days after the first dose and 3 or 7, and 30 days after the second dose.
Arm/Group | Group 3B (V72_41) | Group 3B (V72P10) | Group 3B | Group B_0_1 (V72_41) | Group B_0_1 (V72P10) | Group B_0_1
Number analyzed (Participants) | 144 | 129 | 273 | 105 | 148 | 253
Percentage of subjects
  5/99: number analyzed (Participants) | 134 | 120 | 254 | 100 | 139 | 239
  5/99 | 84 [77 to 90] | 84 [76.4 to 90.2] | 84 [79.2 to 88.5] | 7 [2.9 to 13.9] | 24 [16.9 to 31.7] | 17 [12.2 to 22.1]
  NZ98/254 | 9 [4.9 to 14.9] | 29 [21.1 to 37.3] | 18 [13.9 to 23.4] | 0 [0 to 3.5] | 14 [9 to 20.9] | 8 [5.2 to 12.4]
Statistical Analysis 1: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); The group difference in percentages of subjects with response against N. meningitidis group B indicator strain 5/99 and the associated confidence interval for the difference was calculated using the method of Miettinen and Nurminen; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 [(Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; Miettinen and Nurminen score method; Vaccine Group Difference = 77, 95% CI 2-sided [68.1 to 84.1]
Statistical Analysis 2: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 1, analysis 1]; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 [Group 3B (V72P10) vs. Group B_0_1 (V72P10)]; Miettinen and Nurminen score method; Vaccine group difference = 60, 95% CI 2-sided [49.9 to 69.2]
Statistical Analysis 3: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 1, analysis 1]; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 (Group 3B vs. Group B_0_1); Miettinen and Nurminen score method; Vaccine group difference = 68, 95% CI 2-sided [60.5 to 73.5]
Statistical Analysis 4: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); The group difference in percentages of subjects with response against N. meningitidis group B indicator strain NZ98/254 and the associated confidence interval for the difference was calculated using the method of Miettinen and Nurminen; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 [Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; Miettinen and Nurminen score method; Vaccine group difference = 9, 95% CI 2-sided [5.3 to 14.8]
Statistical Analysis 5: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 1, analysis 4]; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 [Group 3B (V72P10 vs. Group B_0_1 (V72P10)]; Miettinen and Nurminen score method; Vaccine group difference = 14, 95% CI 2-sided [4.9 to 24.2]
Statistical Analysis 6: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 1, analysis 4]; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 (Group 3B vs. Group B_0_1); Miettinen and Nurminen score method; Vaccine group difference = 10, 95% CI 2-sided [4.3 to 15.9]

2. Primary Outcome: Percentage of Subjects With hSBA≥1:5
Description: Bactericidal activity was measured against the N. meningitidis group B indicator strains H44/76 and M10713. This outcome measure was assessed only for strains H44/76 and M10713.
Time Frame: Group 3B: Day 1 (prior to booster dose); Group B_0_1: Day 1 (prior to first dose).
Population: Analysis was performed on the Full analysis set (FAS) persistence.The FAS included all follow-on subjects (Group 3B) in the All Enrolled Set, and all naïve subjects (group B_0_1) in the All Enrolled Set who provided evaluable immunogenicity result at day 1, for at least one indicator strain.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Group 3B (V72_41) | Group 3B (V72P10) | Group 3B | Group B_0_1 (V72_41) | Group B_0_1 (V72P10) | Group B_0_1
Number analyzed (Participants) | 144 | 131 | 275 | 105 | 150 | 255
Percentage of subjects
  H44/76 | 26 [19.4 to 34.4] | 41 [32.7 to 50.2] | 33 [27.9 to 39.4] | 5 [1.6 to 10.8] | 11 [6.7 to 17.5] | 9 [5.5 to 12.8]
  M10713: number analyzed (Participants) | 143 | 131 | 274 | 105 | 150 | 255
  M10713 | 71 [63.2 to 78.6] | 78 [69.8 to 84.6] | 74 [68.9 to 79.5] | 59 [49.0 to 68.5] | 78 [70.5 to 84.3] | 70 [64.2 to 75.7]
Statistical Analysis 1: Comparison: Group 3B vs Group B_0_1; The group difference in percentages of subjects with response against N. meningitidis group B indicator strain H44/76and the associated confidence interval for the difference was calculated using the method of Miettinen and Nurminen; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 (Group 3B vs. Group B_0_1); Miettinen and Nurminen score method; vaccine group difference = 25, 95% CI 2-sided [18.2 to 31.4]
Statistical Analysis 2: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); The group difference in percentages of subjects with response against N. meningitidis group B indicator strain H44/76 and the associated confidence interval for the difference was calculated using the method of Miettinen and Nurminen; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 [(Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; Miettinen and Nurminen score method; Vaccine groups difference = 22, 95% CI 2-sided [13.2 to 30.1]
Statistical Analysis 3: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 2, analysis 2]; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 [Group 3B (V72P10) vs. Group B_0_1 (V72P10)]; Miettinen and Nurminen score method; Vaccine group difference = 30, 95% CI 2-sided [20.0 to 39.6]
Statistical Analysis 4: Comparison: Group 3B vs Group B_0_1; The group difference in percentages of subjects with response against N. meningitidis group B indicator strain M10713 and the associated confidence interval for the difference was calculated using the method of Miettinen and Nurminen; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 (Group 3B vs. Group B_0_1); Miettinen and Nurminen score method; Vaccine group difference = 4, 95% CI 2-sided [-3.4 to 11.9]
Statistical Analysis 5: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 2, analysis 4]; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 [Group 3B (V72_41) vs. Group B_0_1(V72_41)]; Miettinen and Nurminen score method; vaccine group differences = 12, 95% CI 2-sided [0.33 to 24.2]
Statistical Analysis 6: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 2, analysis 4]; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 [Group 3B (V72P10) vs. Group B_0_1(V72P10)]; Miettinen and Nurminen score method; Vaccine group difference = 0, 95% CI 2-sided [-10.0 to 9.5]

3. Primary Outcome: Percentage of Subjects With hSBA Titers≥1:5 in Parent Studies-V72P10 and V72_41
Description: Bactericidal activity was measured against the N. meningitidis group B indicator strains H44/76 and M10713
Time Frame: At one month after last vaccination in parent studies- V72P10 (Month 7) and V72_41 (Month 2)
Population: Analysis was performed on the Full analysis set (FAS) persistence. The FAS included all follow-on subjects (Group 3B) in the All Enrolled Set, and all naïve subjects (group B_0_1) in the All Enrolled Set who provided evaluable immunogenicity result at day 1, for at least one indicator strain.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Group 3B (V72_41) | Group 3B (V72P10)
Number analyzed (Participants) | 144 | 131
Percentage of subjects
  H44/76- Baseline in Parent study | 1 [0.17 to 4.9] | 23 [16 to 31.1]
  H44/76- 1 month after last vacc in Parent study | 99 [95.1 to 99.83] | 100 [97.2 to 100]
  M10713- Baseline in Parent study: number analyzed (Participants) | 143 | 131
  M10713- Baseline in Parent study | 34 [25.9 to 41.9] | 73 [64 to 80]
  M10713- 1 month after last vacc in Parent study: number analyzed (Participants) | 140 | 131
  M10713- 1 month after last vacc in Parent study | 68 [59.4 to 75.5] | 98 [94.6 to 99.81]

4. Primary Outcome: Percentage of Subjects With hSBA≥1:8
Description: Bactericidal activity was measured against each of the N. meningitidis group B indicator strains H44/76,5/99,NZ98/254 and M10713
Time Frame: Group 3B: Day 1 (prior to booster dose); Group B_0_1: Day 1 (prior to first dose).
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Group 3B (V72_41) | Group 3B (V72P10) | Group 3B | Group B_0_1 (V72_41) | Group B_0_1 (V72P10) | Group B_0_1
Number analyzed (Participants) | 144 | 131 | 275 | 105 | 150 | 255
Percentage of subjects
  H44/76 | 22 [15.7 to 29.9] | 35 [27.0 to 43.9] | 28 [23.1 to 34.1] | 1 [0.02 to 5.2] | 9 [5.2 to 15.2] | 6 [3.3 to 9.5]
  5/99: number analyzed (Participants) | 134 | 120 | 254 | 100 | 139 | 239
  5/99 | 78 [70.4 to 85.0] | 83 [75.4 to 89.5] | 81 [75.3 to 85.4] | 4 [1.1 to 9.9] | 19 [13.2 to 27.0] | 13 [9.0 to 17.9]
  NZ98/254: number analyzed (Participants) | 144 | 129 | 273 | 105 | 148 | 253
  NZ98/254 | 7 [3.4 to 12.4] | 22 [15.6 to 30.7] | 14 [10.4 to 19.0] | 0 [0.0 to 3.5] | 9 [5.3 to 15.4] | 6 [3.1 to 9.1]
  M10713: number analyzed (Participants) | 143 | 131 | 274 | 105 | 150 | 255
  M10713 | 62 [53.0 to 69.5] | 75 [66.5 to 82.0] | 68 [62.0 to 73.4] | 52 [42.4 to 62.2] | 71 [62.7 to 77.8] | 63 [56.9 to 69.1]
Statistical Analysis 1: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 2, analysis 2]; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 (Group 3B vs. Group B_0_1); Miettinen and Nurminen score method; Vaccine group difference = 22, 95% CI 2-sided [16.5 to 28.6]
Statistical Analysis 2: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 2, analysis 2]; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 [Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; Miettinen and Nurminen score method; Vaccine group difference = 21, 95% CI 2-sided [14.6 to 28.9]
Statistical Analysis 3: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 2, analysis 1]; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 [Group 3B (V72P10) vs. Group B_0_1 (V72P10)]; Miettinen and Nurminen score method; Vaccine group difference = 26, 95% CI 2-sided [16.4 to 35.3]
Statistical Analysis 4: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 1, analysis 1]; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 (Group 3B vs. Group B_0_1); Miettinen and Nurminen score method; Vaccine group difference = 68, 95% CI 2-sided [60.8 to 73.7]
Statistical Analysis 5: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 1, analysis 1]; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 [Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; Miettinen and Nurminen score method; Vaccine group difference = 74, 95% CI 2-sided [65.3 to 81.3]
Statistical Analysis 6: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 1, analysis 1]; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 [Group 3B (V72P10) vs. Group B_0_1 (V72P10)]; Miettinen and Nurminen score method; Vaccine group difference = 64, 95% CI 2-sided [53.6 to 72.3]
Statistical Analysis 7: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 1, analysis 4]; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 (Group 3B vs. Group B_0_1); Miettinen and Nurminen score method; Vaccine group difference = 9, 95% CI 2-sided [3.7 to 14.0]
Statistical Analysis 8: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 1, analysis 4]; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 [Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; Miettinen and Nurminen score method; Vaccine group difference = 7, 95% CI 2-sided [3.3 to 12.3]
Statistical Analysis 9: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 1, analysis 4]; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 [Group 3B (V72P10) vs. Group B_0_1 (V72P10)]; Miettinen and Nurminen score method; Vaccine group difference = 13, 95% CI 2-sided [4.5 to 22.0]
Statistical Analysis 10: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 2, analysis 4]; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 (Group 3B vs. Group B_0_1); Miettinen and Nurminen score method; Vaccine group difference = 5, 95% CI 2-sided [-3.4 to 12.8]
Statistical Analysis 11: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 2, analysis 4]; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 [Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; Miettinen and Nurminen score method; Vaccine group difference = 9, 95% CI 2-sided [-3.3 to 21.4]
Statistical Analysis 12: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 2, analysis 4]; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 [Group 3B (V72P10) vs. Group B_0_1 (V72P10)]; Miettinen and Nurminen score method; Vaccine group difference = 4, 95% CI 2-sided [-6.4 to 14.5]

5. Primary Outcome: Percentage of Subjects With hSBA≥1:16
Description: as for outcome 4
Time Frame: Group 3B: Day 1 (prior to booster dose); Group B_0_1: Day 1 (prior to first dose).
Population: Analysis was performed on the Full analysis set (FAS) persistence. The FAS included all follow-on subjects (Group 3B) in the All Enrolled Set, and all naïve subjects in the All Enrolled Set who provided evaluable immunogenicity result at day 1, for at least one indicator strain.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Group 3B (V72_41) | Group 3B (V72P10) | Group 3B | Group B_0_1 (V72_41) | Group B_0_1 (V72P10) | Group B_0_1
Number analyzed (Participants) | 144 | 131 | 275 | 105 | 150 | 255
Percentage of subjects
  H44/76 | 12 [7.0 to 18.2] | 28 [20.7 to 36.8] | 20 [15.1 to 24.8] | 0 [0.0 to 3.5] | 7 [3.7 to 12.7] | 4 [2.2 to 7.6]
  5/99: number analyzed (Participants) | 134 | 120 | 254 | 100 | 139 | 239
  5/99 | 72 [63.2 to 79.1] | 78 [69.9 to 85.3] | 75 [69.0 to 80.0] | 2 [0.24 to 7.0] | 13 [7.9 to 19.7] | 8 [5.2 to 12.6]
  NZ98/254: number analyzed (Participants) | 144 | 129 | 273 | 105 | 148 | 253
  NZ98/254 | 5 [2.0 to 9.8] | 19 [12.3 to 26.4] | 11 [7.8 to 15.7] | 0 [0.0 to 3.5] | 4 [1.5 to 8.6] | 2 [0.9 to 5.1]
  M10713: number analyzed (Participants) | 143 | 131 | 274 | 105 | 150 | 255
  M10713 | 50 [41.9 to 58.8] | 65 [56.1 to 73.0] | 57 [51.2 to 63.2] | 48 [37.8 to 57.6] | 61 [53.0 to 69.2] | 56 [49.4 to 61.9]
Statistical Analysis 1: Comparison: Group 3B vs Group B_0_1; The group difference in percentages of subjects with response against N. meningitidis serogroup B indicator strain H44/76 and the associated confidence interval for the difference was calculated using the method of Miettinen and Nurminen; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 (Group 3B vs. Group B_0_1); Miettinen and Nurminen score method; Vaccine group difference = 15, 95% CI 2-sided [10.1 to 20.9]
Statistical Analysis 2: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 5, analysis 1]; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 [Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; Miettinen and Nurminen score method; Vaccine group difference = 12, 95% CI 2-sided [7.5 to 18.1]
Statistical Analysis 3: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 5, analysis 1]; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 [Group 3B (V72P10) vs. Group B_0_1 (V72P10)]; Miettinen and Nurminen score method; Vaccine group difference = 21, 95% CI 2-sided [12.3 to 29.9]
Statistical Analysis 4: Comparison: Group 3B vs Group B_0_1; The group difference in percentages of subjects with response against N. meningitidis serogroup B indicator strain 5/99 and the associated confidence interval for the difference was calculated using the method of Miettinen and Nurminen; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 (Group 3B vs. Group B_0_1); Miettinen and Nurminen score method; vaccine group difference = 66, 95% CI 2-sided [59.6 to 72.4]
Statistical Analysis 5: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 5, analysis 4]; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 [Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; Miettinen and Nurminen score method; Vaccine group difference = 70, 95% CI 2-sided [60.8 to 77.0]
Statistical Analysis 6: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 5, analysis 4]; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 [Group 3B (V72P10) vs. Group B_0_1 (V72P10)]; Miettinen and Nurminen score method; Vaccine group difference = 65, 95% CI 2-sided [55.2 to 73.7]
Statistical Analysis 7: Comparison: Group 3B vs Group B_0_1; The group difference in percentages of subjects with response against N. meningitidis serogroup B indicator strain NZ98/254 and the associated confidence interval for the difference was calculated using the method of Miettinen and Nurminen; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 (Group 3B vs. Group B_0_1); Miettinen and Nurminen score method; Vaccine group difference = 9, 95% CI 2-sided [4.9 to 13.6]
Statistical Analysis 8: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 5, analysis 7]; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 [Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; Miettinen and Nurminen score method; Vaccine group difference = 5, 95% CI 2-sided [1.2 to 9.7]
Statistical Analysis 9: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 5, analysis 7]; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 [Group 3B (V72P10) vs. Group B_0_1 (V72P10)]; Miettinen and Nurminen score method; Vaccine group difference = 15, 95% CI 2-sided [7.5 to 22.6]
Statistical Analysis 10: Comparison: Group 3B vs Group B_0_1; The group difference in percentages of subjects with response against N. meningitidis serogroup B indicator strain M10713 and the associated confidence interval for the difference was calculated using the method of Miettinen and Nurminen; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 (Group 3B vs. Group B_0_1); Miettinen and Nurminen score method; Vaccine group difference = 2, 95% CI 2-sided [-6.8 to 10.0]
Statistical Analysis 11: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 5, analysis 10]; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 [Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; Miettinen and Nurminen score method; Vaccine group difference = 3, 95% CI 2-sided [-9.8 to 15.2]
Statistical Analysis 12: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 5, analysis 10]; Test type: Other — Vaccine comparison at Persistence at 4/7.5 years/Baseline in V72_75 [Group 3B (V72P10) vs. Group B_0_1 (V72P10)]; Miettinen and Nurminen score method; Vaccine group difference = 4, 95% CI 2-sided [-7.8 to 14.7]

6. Primary Outcome: hSBA Geometric Mean Titers (GMTs) After the Last Dose of rMenB+OMV NZ Vaccination in the Parent Study.
Description: Bactericidal activity was measured against each of the N. meningitidis group B indicator strains H44/76,5/99, NZ98/254 a nd M10713.
Time Frame: Group 3B: 1 month after the last rMenB+OMV NZ vaccination in parent study and Day 1(prior to booster dose); Group B_0_1: Day 1(prior to first dose)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 3B (V72_41) | Group 3B (V72P10) | Group 3B | Group B_0_1 (V72_41) | Group B_0_1 (V72P10) | Group B_0_1
Number analyzed (Participants) | 144 | 131 | 275 | 105 | 150 | 255
Titers
  H44/76(1 month post last vacc in parent study): number analyzed (Participants) | 144 | 131 | 275 | 0 | 0 | 0
  H44/76(1 month post last vacc in parent study) | 99 [82 to 119] | 197 [165 to 235] | 124 [108 to 143] |  |  |
  H44/76( Day 1) | 2.43 [2.04 to 2.89] | 4.51 [3.57 to 5.69] | 3.05 [2.61 to 3.56] | 1.14 [0.93 to 1.40] | 1.52 [1.23 to 1.90] | 1.20 [1.02 to 1.42]
  5/99(1 month post last vacc in parent study): number analyzed (Participants) | 134 | 120 | 254 | 0 | 0 | 0
  5/99(1 month post last vacc in parent study) | 180 [153 to 211] | 606 [492 to 746] | 270 [234 to 311] |  |  |
  5/99 (Day 1): number analyzed (Participants) | 134 | 120 | 254 | 100 | 139 | 239
  5/99 (Day 1) | 24 [19 to 30] | 31 [23 to 42] | 26 [21 to 31] | 1.20 [0.91 to 1.58] | 2.30 [1.75 to 3.04] | 1.57 [1.26 to 1.95]
  NZ98/254(1 month post last vacc in parent study): number analyzed (Participants) | 144 | 129 | 273 | 0 | 0 | 0
  NZ98/254(1 month post last vacc in parent study) | 11 [8.67 to 14] | 93 [75 to 117] | 22 [19 to 27] |  |  |
  NZ98/254( Day 1): number analyzed (Participants) | 144 | 129 | 273 | 105 | 148 | 253
  NZ98/254( Day 1) | 1.31 [1.17 to 1.45] | 2.56 [2.07 to 3.17] | 1.66 [1.46 to 1.89] | 1.01 [0.89 to 1.14] | 1.50 [1.23 to 1.84] | 1.11 [0.97 to 1.27]
  M10713(1 month post last vacc in parent study): number analyzed (Participants) | 140 | 131 | 271 | 0 | 0 | 0
  M10713(1 month post last vacc in parent study) | 10 [7.65 to 14] | 66 [53 to 81] | 19 [16 to 24] |  |  |
  M10713(Day 1): number analyzed (Participants) | 140 | 131 | 271 | 105 | 150 | 255
  M10713(Day 1) | 13 [9.86 to 18] | 22 [16 to 29] | 16 [13 to 20] | 10 [7.13 to 15] | 18 [14 to 24] | 12 [9.86 to 16]
Statistical Analysis 1: Comparison: Group 3B vs Group B_0_1; Adjusted geometric mean titers for H44/76 indicator strain were obtained by exponentiating (base 10) the least square means and the lower and upper limits of the 95% confidence intervals of the log-transformed titers obtained from an ANOVA estimation adjusting for vaccine group and country; Test type: Other — Vaccine Comparison at Persistence at 4 years/Baseline in V72_75 (Group 3B vs. Group B_0_1); ANOVA; Adjusted by vaccine group and country; vaccine group ratio of GMTs = 2.54, 95% CI 2-sided [2.07 to 3.12]
Statistical Analysis 2: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 6, analysis 1]; Test type: Other — Vaccine Comparison at Persistence at 4 years/Baseline in V72_75 [Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; ANOVA; Adjusted by vaccine group and country; vaccine group ratio of GMTs = 2.13, 95% CI 2-sided [1.66 to 2.72]
Statistical Analysis 3: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 6, analysis 1]; Test type: Other — Vaccine Comparison at Persistence at 4 years/Baseline in V72_75 [Group 3B (V72P10) vs. Group B_0_1 (V72P10)]; ANOVA; Adjusted by vaccine group and country; vaccine group ratio of GMTs = 2.96, 95% CI 2-sided [2.15 to 4.07]
Statistical Analysis 4: Comparison: Group 3B vs Group B_0_1; Adjusted geometric mean titers for 5/99 indicator strain were obtained by exponentiating (base 10) the least square means and the lower and upper limits of the 95% confidence intervals of the log-transformed titers obtained from an ANOVA estimation adjusting for vaccine group and country; Test type: Other — Vaccine Comparison at Persistence at 4 years/Baseline in V72_75 (Group 3B vs. Group B_0_1); ANOVA; Adjusted by vaccine group and country; Vaccine group ratio of GMTs = 16, 95% CI 2-sided [12 to 21]
Statistical Analysis 5: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 6, analysis 4]; Test type: Other — Vaccine Comparison at Persistence at 4 years/Baseline in V72_75 [Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; ANOVA; Adjusted by vaccine group and country; vaccine group ratio of GMTs = 20, 95% CI 2-sided [14 to 28]
Statistical Analysis 6: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 6, analysis 4]; Test type: Other — Vaccine Comparison at Persistence at 4 years/Baseline in V72_75 [Group 3B (V72P10) vs. Group B_0_1 (V72P10)]; ANOVA; Adjusted by vaccine group and country; vaccine group ratio of GMTs = 14, 95% CI 2-sided [9.05 to 20]
Statistical Analysis 7: Comparison: Group 3B vs Group B_0_1; Adjusted geometric mean titers for NZ98/254 indicator strain were obtained by exponentiating (base 10) the least square means and the lower and upper limits of the 95% confidence intervals of the log-transformed titers obtained from an ANOVA estimation adjusting for vaccine group and country; Test type: Other — Vaccine Comparison at Persistence at 4 years/Baseline in V72_75 (Group 3B vs. Group B_0_1); ANOVA; Adjusted by vaccine group and country; Vaccine group ratio of GMTs = 1.50, 95% CI 2-sided [1.26 to 1.78]
Statistical Analysis 8: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 6, analysis 7]; Test type: Other — Vaccine Comparison at Persistence at 4 years/Baseline in V72_75 [Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; ANOVA; Adjusted by vaccine group and country; vaccine group ratio of GMTs = 1.30, 95% CI 2-sided [1.11 to 1.51]
Statistical Analysis 9: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 6, analysis 7]; Test type: Other — Vaccine Comparison at Persistence at 4 years/Baseline in V72_75 [Group 3B (V72P10) vs. Group B_0_1 (V72P10)]; ANOVA; Adjusted by vaccine group and country; vaccine group ratio of GMTs = 1.70, 95% CI 2-sided [1.27 to 2.28]
Statistical Analysis 10: Comparison: Group 3B vs Group B_0_1; Adjusted geometric mean titers for M10713 indicator strain were obtained by exponentiating (base 10) the least square means and the lower and upper limits of the 95% confidence intervals of the log-transformed titers obtained from an ANOVA estimation adjusting for vaccine group and country; Test type: Other — Vaccine Comparison at Persistence at 4 years/Baseline in V72_75 (Group 3B vs. Group B_0_1); ANOVA; Adjusted by vaccine group and country; Vaccine group ratio of GMTs = 1.26, 95% CI 2-sided [0.94 to 1.68]
Statistical Analysis 11: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 6, analysis 10]; Test type: Other — Vaccine Comparison at Persistence at 4 years/Baseline in V72_75 [Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; ANOVA; Adjusted by vaccine group and country; vaccine group ratio of GMTs = 1.32, 95% CI 2-sided [0.85 to 2.05]
Statistical Analysis 12: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 6, analysis 10]; Test type: Other — Vaccine Comparison at Persistence at 4 years/Baseline in V72_75 [Group 3B (V72P10) vs. Group B_0_1 (V72P10)]; ANOVA; Adjusted by vaccine group and country; vaccine group ratio of GMTs = 1.20, 95% CI 2-sided [0.81 to 1.78]

7. Primary Outcome: Geometric Mean Ratios (GMRs) of GMTs After the Last Dose of rMenB+OMV NZ Vaccination in the Parent Study Versus Day 1.
Description: The GMRs of GMTs at Day 1 versus one month after the last dose of rMenB+OMV NZ vaccination in the parent study were calculated. Bactericidal activity was measured against each of the N. meningitidis group B indicator strains H44/76, 5/99,NZ98/254 and M10713.
Time Frame: Group 3B: 1 month after the last vaccination in parent study and Day 1 (prior to booster dose)
Population: Analysis was performed on the Full analysis set (FAS) persistence. The FAS included all follow-on subjects (Group 3B) in the All Enrolled Set, and all naïve subjects (B_0_1) in the All Enrolled Set who provided evaluable immunogenicity result at day 1, for at least one indicator strain.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Group 3B (V72_41) | Group 3B (V72P10) | Group 3B
Number analyzed (Participants) | 144 | 131 | 275
Ratio
  H44/76 | 0.026 [0.020 to 0.033] | 0.023 [0.018 to 0.029] | 0.025 [0.020 to 0.030]
  5/99: number analyzed (Participants) | 134 | 120 | 254
  5/99 | 0.13 [0.10 to 0.18] | 0.052 [0.039 to 0.068] | 0.098 [0.079 to 0.12]
  NZ98/254: number analyzed (Participants) | 144 | 129 | 273
  NZ98/254 | 0.12 [0.092 to 0.15] | 0.027 [0.021 to 0.036] | 0.073 [0.059 to 0.089]
  M10713: number analyzed (Participants) | 140 | 131 | 271
  M10713 | 1.26 [0.92 to 1.73] | 0.33 [0.25 to 0.43] | 0.81 [0.65 to 1.01]

8. Primary Outcome: Number of Subjects With Solicited Local and Systemic AEs.
Description: Solicited adverse events are signs and symptoms derived from organized data collection systems, such as Subject Diaries or interview. The percentage and frequencies of subjects reporting solicited local and systemic AEs were tabulated. Threshold for any Erythema, Swelling and Induration: >= 25 mm Note:Vaccination 2 was performed only on group B_0_1 subjects. Threshold for any Erythema, Swelling and Induration: >= 25 mm
Time Frame: 7 days (including the day of vaccination) after each vaccination
Population: The analysis was done on the Solicited Safety Set. The solicited safety set included all subjects in the exposed set with any solicited adverse event data and/indicators of solicited adverse events.
Measure: Number; unit: Subjects
Arm/Group | Group 3B | Group B_0_1
Number analyzed (Participants) | 266 | 254
Subjects
  Any | 263 | 251
  Any Local (vaccination 1): number analyzed (Participants) | 266 | 253
  Any Local (vaccination 1) | 258 | 247
  Injection site pain (vaccination 1): number analyzed (Participants) | 264 | 252
  Injection site pain (vaccination 1) | 258 | 247
  Erythema (vaccination 1): number analyzed (Participants) | 261 | 248
  Erythema (vaccination 1) | 54 | 18
  Swelling (vaccination 1): number analyzed (Participants) | 261 | 249
  Swelling (vaccination 1) | 60 | 34
  Induration (vaccination 1): number analyzed (Participants) | 261 | 248
  Induration (vaccination 1) | 54 | 26
  Any systemic (vaccination 1): number analyzed (Participants) | 266 | 253
  Any systemic (vaccination 1) | 203 | 163
  Fever (≥ 38.0°C) (vaccination 1): number analyzed (Participants) | 265 | 253
  Fever (≥ 38.0°C) (vaccination 1) | 16 | 4
  High fever (≥ 39.5°C) (vaccination 1): number analyzed (Participants) | 265 | 253
  High fever (≥ 39.5°C) (vaccination 1) | 0 | 0
  Nausea (vaccination 1): number analyzed (Participants) | 264 | 252
  Nausea (vaccination 1) | 56 | 30
  Fatigue (vaccination 1): number analyzed (Participants) | 266 | 252
  Fatigue (vaccination 1) | 155 | 110
  Myalgia (vaccination 1): number analyzed (Participants) | 265 | 252
  Myalgia (vaccination 1) | 120 | 71
  Arthralgia (vaccination 1): number analyzed (Participants) | 265 | 252
  Arthralgia (vaccination 1) | 84 | 47
  Headache (vaccination 1): number analyzed (Participants) | 266 | 253
  Headache (vaccination 1) | 146 | 94
  Any Local (vaccination 2): number analyzed (Participants) | 0 | 248
  Any Local (vaccination 2) |  | 226
  Injection site pain (vaccination 2): number analyzed (Participants) | 0 | 247
  Injection site pain (vaccination 2) |  | 226
  Erythema (vaccination 2): number analyzed (Participants) | 0 | 247
  Erythema (vaccination 2) |  | 21
  Swelling (vaccination 2): number analyzed (Participants) | 0 | 248
  Swelling (vaccination 2) |  | 32
  Induration (vaccination 2): number analyzed (Participants) | 0 | 247
  Induration (vaccination 2) |  | 31
  Any systemic (vaccination 2): number analyzed (Participants) | 0 | 248
  Any systemic (vaccination 2) |  | 140
  Fever (≥ 38.0°C) (vaccination 2): number analyzed (Participants) | 0 | 248
  Fever (≥ 38.0°C) (vaccination 2) |  | 5
  High fever (≥ 39.5°C) (vaccination 2): number analyzed (Participants) | 0 | 248
  High fever (≥ 39.5°C) (vaccination 2) |  | 0
  Nausea (vaccination 2): number analyzed (Participants) | 0 | 248
  Nausea (vaccination 2) |  | 33
  Fatigue (vaccination 2): number analyzed (Participants) | 0 | 248
  Fatigue (vaccination 2) |  | 92
  Myalgia (vaccination 2): number analyzed (Participants) | 0 | 248
  Myalgia (vaccination 2) |  | 64
  Arthralgia (vaccination 2): number analyzed (Participants) | 0 | 248
  Arthralgia (vaccination 2) |  | 36
  Headache (vaccination 2): number analyzed (Participants) | 0 | 248
  Headache (vaccination 2) |  | 84

9. Primary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs).
Description: An unsolicited adverse event is an adverse event that was not solicited using a subject Diary and that was spontaneously communicated by a subject and/or parent(s)/legal guardian(s) who has signed the informed consent. Note : Vaccination 2 was performed only on group B_0_1 subjects.
Time Frame: 30 days (including the day of vaccination) after each vaccination.
Population: Analysis was performed on the unsolicited safety set. The unsolicited safety set included all subjects who received a study vaccination with unsolicited adverse event data.
Measure: Number; unit: Subjects
Arm/Group | Group 3B | Group B_0_1
Number analyzed (Participants) | 275 | 255
Subjects
  Any | 87 | 131
  Any unsolicited AEs ( vaccination 1) | 87 | 96
  Any unsolicited AEs (vaccination 2): number analyzed (Participants) | 0 | 250
  Any unsolicited AEs (vaccination 2) |  | 73

10. Primary Outcome: Number of Subjects With Any SAEs, AEs Leading to Withdrawal and Medically Attended AEs.
Description: A serious adverse event is any untoward medical occurrence that at any dose results in death or is life threatening or requires prolonged hospitalization, leads to Persistent or significant disability/incapacity.
Time Frame: Group 3B: from Day 1 to Day 31 (study termination visit) and Group B_0_1: from Day 1 to Day 61 (study termination visit)
Population: Analysis was performed on the Overall safety set. The overall safety set included all screened subjects in the solicited and unsolicited safety set who provided informed consent and provided demographic and/or baseline screening assessments, regardless of the subject's randomization and treatment status in the study and received a Subject ID.
Measure: Number; unit: Subjects
Arm/Group | Group 3B | Group B_0_1
Number analyzed (Participants) | 275 | 255
Subjects
  Any SAEs | 0 | 1
  Any Medically Attended AEs | 17 | 34
  Any AEs leading to premature withdrawal | 0 | 1

11. Secondary Outcome: Percentage of Subjects With hSBA ≥1:4 After Booster Dose/First Vaccination of rMenB+OMV NZ.
Description: as for outcome 1
Time Frame: Group 3B: 30 days after booster dose, Group B_0_1 : 30 days after first vaccination.
Population: Analysis was performed on the Full Analysis set( FAS) booster. The FAS booster included all follow on subjects and all naive subjects in the All enrolled set who received vaccination at day 1 and provided evaluable immunogenicity result at day 31 for at least one indicator strain.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Group 3B (V72_41) | Group 3B (V72P10) | Group 3B | Group B_0_1 (V72_41) | Group B_0_1 (V72P10) | Group B_0_1
Number analyzed (Participants) | 142 | 120 | 262 | 103 | 148 | 251
Percentage of subjects
  5/99: number analyzed (Participants) | 124 | 102 | 226 | 97 | 137 | 234
  5/99 | 100 [97.1 to 100.0] | 100 [96.4 to 100.0] | 100 [98.4 to 100.0] | 87 [78.2 to 92.7] | 84 [76.7 to 89.7] | 85 [79.8 to 89.4]
  NZ98/254 | 94 [89.2 to 97.5] | 93 [87.3 to 97.1] | 94 [90.3 to 96.5] | 41 [31.2 to 50.9] | 62 [53.8 to 70.0] | 53 [47.0 to 59.7]
Statistical Analysis 1: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); The group difference in percentages of subjects with response against N. meningitidis serogroup B indicator strain 5/99 and the associated confidence interval for the difference were calculated using the method of Miettinen and Nurminen; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 [Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; Miettinen and Nurminen score method; Vaccine group difference = 13, 95% CI 2-sided [8.0 to 21.6]
Statistical Analysis 2: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 11, analysis 1]; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 [Group 3B (V72P10) vs. Group B_0_1 (V72P10)]; Miettinen and Nurminen score method; Vaccine group difference = 16, 95% CI 2-sided [10.8 to 23.1]
Statistical Analysis 3: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 11, analysis 1]; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 (Group 3B vs. Group B_0_1); Miettinen and Nurminen score method; Vaccine group difference = 15, 95% CI 2-sided [11.0 to 20.1]
Statistical Analysis 4: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); The group difference in percentages of subjects with response against N. meningitidis serogroup B indicator strain NZ98/254 and the associated confidence interval for the difference were calculated using the method of Miettinen and Nurminen; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 [Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; Miettinen and Nurminen score method; Vaccine group difference = 54, 95% CI 2-sided [43.0 to 63.3]
Statistical Analysis 5: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 11, analysis 4]; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 [Group 3B (V72P10) vs. Group B_0_1 (V72P10)]; Miettinen and Nurminen score method; Vaccine group difference = 31, 95% CI 2-sided [22.0 to 40.1]
Statistical Analysis 6: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 11, analysis 4]; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 (Group 3B vs. Group B_0_1); Miettinen and Nurminen score method; Vaccine group difference = 41, 95% CI 2-sided [33.6 to 47.2]

12. Secondary Outcome: Percentage of Subjects With hSBA ≥1:5 After Booster Dose/First Vaccination of rMenB+OMV NZ.
Description: as for outcome 2
Time Frame: Group 3B: 30 days after booster dose, Group B_0_1 : 30 days after first vaccination.
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Group 3B (V72_41) | Group 3B (V72P10) | Group 3B | Group B_0_1 (V72_41) | Group B_0_1 (V72P10) | Group B_0_1
Number analyzed (Participants) | 141 | 127 | 268 | 104 | 149 | 253
Percentage of subjects
  H44/76 | 98 [93.9 to 99.56] | 100 [97.1 to 100.0] | 99 [96.8 to 99.77] | 80 [70.8 to 87.0] | 79 [71.1 to 84.8] | 79 [73.5 to 83.9]
  M10713: number analyzed (Participants) | 141 | 127 | 268 | 103 | 149 | 252
  M10713 | 99 [96.1 to 99.98] | 98 [94.4 to 99.81] | 99 [96.8 to 99.77] | 80 [70.5 to 86.9] | 92 [86.4 to 95.8] | 87 [82.1 to 90.8]
Statistical Analysis 1: Comparison: Group 3B vs Group B_0_1; The group difference in percentages of subjects with response against N. meningitidis serogroup B indicator strain H44/76 and the associated confidence interval for the difference were calculated using the method of Miettinen and Nurminen; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 (Group 3B vs. Group B_0_1); Miettinen and Nurminen score method; Vaccine group difference = 20, 95% CI 2-sided [15.0 to 25.4]
Statistical Analysis 2: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 12, analysis 1]; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 [Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; Miettinen and Nurminen score method; Vaccine group difference = 18, 95% CI 2-sided [10.7 to 27.0]
Statistical Analysis 3: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 12, analysis 1]; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 [Group 3B (V72P10) vs. Group B_0_1 (V72P10)]; Miettinen and Nurminen score method; Vaccine group difference = 21, 95% CI 2-sided [15.6 to 28.8]
Statistical Analysis 4: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 5, analysis 10]; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 (Group 3B vs. Group B_0_1); Miettinen and Nurminen score method; vaccine group difference = 12, 95% CI 2-sided [8.0 to 16.8]
Statistical Analysis 5: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 5, analysis 10]; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 [Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; Miettinen and Nurminen score method; Vaccine group difference = 20, 95% CI 2-sided [12.8 to 28.6]
Statistical Analysis 6: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 5, analysis 10]; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 [Group 3B (V72P10) vs. Group B_0_1 (V72P10)]; Miettinen and Nurminen score method; Vaccine group difference = 6, 95% CI 2-sided [1.5 to 12.2]

13. Secondary Outcome: Percentage of Subjects With hSBA ≥1:8 After Booster Dose/First Vaccination of rMenB+OMV NZ
Description: Bactericidal activity was measured against each of the four N. meningitidis group B indicator strains H44/76,5/99,NZ98/254 and M10713.
Time Frame: Group 3B : 30 days after booster dose, Group B_0_1 : 30 days after first vaccination.
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Group 3B (V72_41) | Group 3B (V72P10) | Group 3B | Group B_0_1 (V72_41) | Group B_0_1 (V72P10) | Group B_0_1
Number analyzed (Participants) | 142 | 127 | 268 | 104 | 149 | 253
Percentage of subjects
  H44/76: number analyzed (Participants) | 141 | 127 | 268 | 104 | 149 | 253
  H44/76 | 98 [93.9 to 99.56] | 100 [97.1 to 100.0] | 99 [96.8 to 99.77] | 67 [57.4 to 76.2] | 74 [66.7 to 81.3] | 72 [65.6 to 77.0]
  5/99: number analyzed (Participants) | 124 | 102 | 226 | 97 | 137 | 234
  5/99 | 100 [97.1 to 100] | 100 [96.4 to 100] | 100 [98.4 to 100.0] | 81 [72.3 to 88.6] | 81 [73.4 to 87.2] | 81 [75.6 to 86.0]
  NZ98/254: number analyzed (Participants) | 142 | 120 | 262 | 103 | 148 | 251
  NZ98/254 | 86 [79.1 to 91.2] | 89 [82.2 to 94.1] | 87 [82.8 to 91.2] | 28 [19.7 to 37.9] | 56 [47.7 to 64.2] | 45 [38.4 to 51.0]
  M10713: number analyzed (Participants) | 141 | 127 | 268 | 103 | 149 | 252
  M10713 | 99 [95.0 to 99.83] | 98 [93.3 to 99.51] | 98 [95.7 to 99.4] | 79 [69.5 to 86.1] | 89 [83.1 to 93.7] | 85 [79.9 to 89.1]
Statistical Analysis 1: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 12, analysis 1]; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 (Group 3B vs. Group B_0_1); Miettinen and Nurminen score method; Vaccine group difference = 27, 95% CI 2-sided [21.9 to 33.3]
Statistical Analysis 2: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 12, analysis 1]; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 [Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; Miettinen and Nurminen score method; Vaccine group difference = 31, 95% CI 2-sided [21.8 to 40.3]
Statistical Analysis 3: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 12, analysis 1]; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 [Group 3B (V72P10) vs. Group B_0_1 (V72P10)]; Miettinen and Nurminen score method; Vaccine group difference = 26, 95% CI 2-sided [19.2 to 33.1]
Statistical Analysis 4: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 11, analysis 1]; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 (Group 3B vs. Group B_0_1); Miettinen and Nurminen score method; vaccine group difference = 19, 95% CI 2-sided [14.3 to 24.3]
Statistical Analysis 5: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 11, analysis 1]; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 [Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; Miettinen and Nurminen score method; Vaccine group difference = 19, 95% CI 2-sided [12.1 to 27.5]
Statistical Analysis 6: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 11, analysis 1]; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 [Group 3B (V72P10) vs. Group B_0_1 (V72P10)]; Miettinen and Nurminen score method; Vaccine group difference = 19, 95% CI 2-sided [13.3 to 26.4]
Statistical Analysis 7: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 11, analysis 4]; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 (Group 3B vs. Group B_0_1); Miettinen and Nurminen score method; vaccine group difference = 43, 95% CI 2-sided [35.2 to 49.9]
Statistical Analysis 8: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 11, analysis 4]; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 [Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; Miettinen and Nurminen score method; Vaccine group difference = 58, 95% CI 2-sided [46.6 to 67.3]
Statistical Analysis 9: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 11, analysis 4]; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 [Group 3B (V72P10) vs. Group B_0_1 (V72P10)]; Miettinen and Nurminen score method; Vaccine group difference = 33, 95% CI 2-sided [23.0 to 42.5]
Statistical Analysis 10: Comparison: Group 3B vs Group B_0_1; The group difference in percentages of subjects with response against N. meningitidis serogroup B indicator strain M10713 and the associated confidence interval for the difference were calculated using the method of Miettinen and Nurminen; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 (Group 3B vs. Group B_0_1); Miettinen and Nurminen score method; vaccine group difference = 13, 95% CI 2-sided [8.8 to 18.3]
Statistical Analysis 11: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 13, analysis 10]; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 [Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; Miettinen and Nurminen score method; Vaccine group difference = 20, 95% CI 2-sided [12.6 to 29.0]
Statistical Analysis 12: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 13, analysis 10]; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 [Group 3B (V72P10) vs. Group B_0_1 (V72P10)]; Miettinen and Nurminen score method; Vaccine group difference = 8, 95% CI 2-sided [2.7 to 14.7]

14. Secondary Outcome: Percentage of Subjects With hSBA ≥1:16 After Booster Dose/First Vaccination of rMenB+OMV NZ
Description: Bactericidal activity was measured against each of the four N. meningitidis group B indicator strains H44/76, 5/99, NZ98/254 & M10713.
Time Frame: Group 3B: 30 days after booster dose, Group B_0_1 : 30 days after first vaccination.
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Group 3B (V72_41) | Group 3B (V72P10) | Group 3B | Group B_0_1 (V72_41) | Group B_0_1 (V72P10) | Group B_0_1
Number analyzed (Participants) | 142 | 127 | 268 | 104 | 149 | 253
Percentage of subjects
  H44/76: number analyzed (Participants) | 141 | 127 | 268 | 104 | 149 | 253
  H44/76 | 98 [93.9 to 99.56] | 99 [95.7 to 99.98] | 99 [96.2 to 99.59] | 49 [39.1 to 59.0] | 65 [56.9 to 72.7] | 58 [52.2 to 64.6]
  5/99: number analyzed (Participants) | 124 | 102 | 226 | 97 | 137 | 234
  5/99 | 100 [97.1 to 100] | 100 [96.4 to 100] | 100 [98.4 to 100.0] | 77 [67.7 to 85.2] | 70 [61.7 to 77.6] | 73 [66.9 to 78.6]
  NZ98/254: number analyzed (Participants) | 142 | 120 | 262 | 103 | 148 | 251
  NZ98/254 | 73 [65.2 to 80.3] | 86 [78.3 to 91.5] | 79 [73.6 to 83.8] | 22 [14.7 to 31.6] | 45 [37.1 to 53.7] | 36 [29.9 to 42.1]
  M10713: number analyzed (Participants) | 141 | 127 | 268 | 103 | 149 | 252
  M10713 | 94 [88.2 to 97.0] | 97 [92.1 to 99.1] | 95 [91.8 to 97.4] | 66 [56.0 to 75.1] | 84 [77.0 to 89.4] | 77 [70.9 to 81.7]
Statistical Analysis 1: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 5, analysis 1]; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 (Group 3B vs. Group B_0_1); Miettinen and Nurminen score method; vaccine group difference = 40, 95% CI 2-sided [33.9 to 46.3]
Statistical Analysis 2: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 5, analysis 1]; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 [Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; Miettinen and Nurminen score method; Vaccine group difference = 49, 95% CI 2-sided [38.9 to 58.5]
Statistical Analysis 3: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 5, analysis 1]; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 [Group 3B (V72P10) vs. Group B_0_1 (V72P10)]; Miettinen and Nurminen score method; Vaccine group difference = 34, 95% CI 2-sided [26.6 to 42.2]
Statistical Analysis 4: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 5, analysis 4]; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 (Group 3B vs. Group B_0_1); Miettinen and Nurminen score method; vaccine group difference = 27, 95% CI 2-sided [21.6 to 33.0]
Statistical Analysis 5: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 5, analysis 4]; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 [Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; Miettinen and Nurminen score method; Vaccine group difference = 23, 95% CI 2-sided [15.5 to 32.0]
Statistical Analysis 6: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 5, analysis 4]; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 [Group 3B (V72P10) vs. Group B_0_1 (V72P10)]; Miettinen and Nurminen score method; Vaccine group difference = 30, 95% CI 2-sided [22.9 to 38.1]
Statistical Analysis 7: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 5, analysis 7]; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 (Group 3B vs. Group B_0_1); Miettinen and Nurminen score method; vaccine group difference = 43, 95% CI 2-sided [35.1 to 50.6]
Statistical Analysis 8: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 5, analysis 7]; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 [Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; Miettinen and Nurminen score method; Vaccine group difference = 51, 95% CI 2-sided [39.3 to 60.9]
Statistical Analysis 9: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 5, analysis 7]; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 [Group 3B (V72P10) vs. Group B_0_1 (V72P10)]; Miettinen and Nurminen score method; Vaccine group difference = 41, 95% CI 2-sided [29.9 to 50.2]
Statistical Analysis 10: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 5, analysis 10]; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 (Group 3B vs. Group B_0_1); Miettinen and Nurminen score method; vaccine group difference = 19, 95% CI 2-sided [12.9 to 24.6]
Statistical Analysis 11: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 5, analysis 10]; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 [Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; Miettinen and Nurminen score method; Vaccine group difference = 28, 95% CI 2-sided [17.9 to 37.8]
Statistical Analysis 12: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 5, analysis 10]; Test type: Other — Vaccine comparison at 1 month after booster /1st dose in V72_75 [Group 3B (V72P10) vs. Group B_0_1 (V72P10)]; Miettinen and Nurminen score method; Vaccine group difference = 13, 95% CI 2-sided [6.4 to 20.1]

15. Secondary Outcome: hSBA Geometric Mean Titers Prior to Booster/First Dose of Vaccination & Post Booster/First Dose of Vaccination.
Description: Bactericidal activity was measured against each of the four N. meningitidis group B indicator strains H44/76, 5/99,NZ98/254 and M10713.
Time Frame: Group 3B subjects: Day 1(pre-booster dose) and 30 days post-booster dose. Group B_0_1: Day 1 (pre-first dose) and 30 days post-first dose.
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 3B (V72_41) | Group 3B (V72P10) | Group 3B | Group B_0_1 (V72_41) | Group B_0_1 (V72P10) | Group B_0_1
Number analyzed (Participants) | 142 | 127 | 268 | 104 | 149 | 253
Titers
  H44/76- pre booster/ pre first dose: number analyzed (Participants) | 141 | 127 | 268 | 104 | 149 | 253
  H44/76- pre booster/ pre first dose | 2.45 [2.06 to 2.92] | 4.65 [3.66 to 5.89] | 3.10 [2.65 to 3.62] | 1.13 [0.92 to 1.38] | 1.53 [1.23 to 1.90] | 1.19 [1.01 to 1.41]
  H44/76-1 month post booster/first dose: number analyzed (Participants) | 141 | 127 | 268 | 104 | 149 | 253
  H44/76-1 month post booster/first dose | 158 [123 to 204] | 269 [206 to 351] | 188 [155 to 228] | 13 [10 to 18] | 24 [19 to 31] | 16 [13 to 20]
  5/99- pre booster/ pre first dose: number analyzed (Participants) | 118 | 93 | 211 | 96 | 129 | 225
  5/99- pre booster/ pre first dose | 22 [17 to 28] | 31 [22 to 43] | 24 [19 to 30] | 1.19 [0.89 to 1.59] | 2.19 [1.65 to 2.92] | 1.51 [1.21 to 1.88]
  5/99-1 month post booster/first dose: number analyzed (Participants) | 124 | 102 | 226 | 97 | 137 | 234
  5/99-1 month post booster/first dose | 2191 [1681 to 2856] | 1951 [1425 to 2671] | 2089 [1690 to 2582] | 30 [22 to 40] | 31 [24 to 41] | 31 [25 to 38]
  NZ98/254-pre booster/ pre first dose: number analyzed (Participants) | 142 | 118 | 260 | 103 | 146 | 249
  NZ98/254-pre booster/ pre first dose | 1.31 [1.18 to 1.46] | 2.48 [1.99 to 3.09] | 1.64 [1.44 to 1.86] | 1.00 [0.88 to 1.13] | 1.51 [1.24 to 1.84] | 1.11 [0.97 to 1.28]
  NZ98/254-1 month post booster/first dose: number analyzed (Participants) | 142 | 120 | 262 | 103 | 148 | 251
  NZ98/254-1 month post booster/first dose | 30 [23 to 38] | 41 [30 to 56] | 32 [26 to 39] | 3.58 [2.70 to 4.76] | 9.43 [7.15 to 12] | 5.39 [4.33 to 6.72]
  M10713-pre booster/ pre first dose: number analyzed (Participants) | 140 | 127 | 267 | 103 | 149 | 252
  M10713-pre booster/ pre first dose | 14 [10 to 19] | 22 [16 to 29] | 16 [13 to 20] | 9.82 [6.87 to 14] | 18 [14 to 23] | 12 [9.62 to 15]
  M10713-1 month post booster/first dose: number analyzed (Participants) | 141 | 127 | 268 | 103 | 149 | 252
  M10713-1 month post booster/first dose | 65 [52 to 81] | 113 [90 to 142] | 78 [66 to 92] | 23 [18 to 30] | 46 [37 to 57] | 30 [25 to 36]
Statistical Analysis 1: Comparison: Group 3B vs Group B_0_1; Pre booster/Pre first dose-Adjusted geometric mean titers for H44/76 indicator strain were obtained by exponentiating (base 10) the least square means and the lower and upper limits of the 95% confidence intervals of the log-transformed titers obtained from an ANOVA estimation adjusting for vaccine group and country; Test type: Other — Vaccine comparison Pre-booster or pre-1st dose in V72_75 (Group 3B vs. Group B _0_1); ANOVA; Ratio of GMTs = 2.60, 95% CI 2-sided [2.11 to 3.20]
Statistical Analysis 2: Comparison: Group 3B vs Group B_0_1; Post booster/Post first dose-Adjusted geometric mean titers for H44/76 indicator strain were obtained by exponentiating (base 10) the least square means and the lower and upper limits of the 95% confidence intervals of the log-transformed titers obtained from an ANOVA estimation adjusting for vaccine group and country; Test type: Other — Vaccine comparison Post-booster or post-1st dose in V72_75 (Group 3B vs. Group B _0_1); ANOVA; Ratio of GMTs = 11, 95% CI 2-sided [8.85 to 15]
Statistical Analysis 3: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 15, analysis 1]; Test type: Other — Vaccine comparison-Pre-booster or pre-1st dose in V72_75 [Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; ANOVA; Ratio of GMTs = 2.18, 95% CI 2-sided [1.70 to 2.79]
Statistical Analysis 4: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 15, analysis 2]; Test type: Other — Vaccine comparison-post-booster or post-1st dose in V72_75 [Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; ANOVA; Ratio of GMTs = 12, 95% CI 2-sided [8.22 to 17]
Statistical Analysis 5: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 15, analysis 1]; Test type: Other — Vaccine comparison- Pre-booster or pre-1st dose in V72_75 [Group 3B (V72P10) vs. Group B_0_1 (V72P10)]; ANOVA; Ratio of GMTs = 3.04, 95% CI 2-sided [2.20 to 4.20]
Statistical Analysis 6: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 15, analysis 2]; Test type: Other — Vaccine comparison- post-booster or post-1st dose in V72_75 [Group 3B (V72P10) vs. Group B_0_1 (V72P10)]; ANOVA; Ratio of GMTs = 11, 95% CI 2-sided [7.75 to 16]
Statistical Analysis 7: Comparison: Group 3B vs Group B_0_1; Pre booster/Pre first dose-Adjusted geometric mean titers for 5/99 indicator strain were obtained by exponentiating (base 10) the least square means and the lower and upper limits of the 95% confidence intervals of the log-transformed titers obtained from an ANOVA estimation adjusting for vaccine group and country; Test type: Other — Vaccine comparison Pre-booster or pre-1st dose in V72_75 (Group 3B vs. Group B _0_1); ANOVA; Ratio of GMTs = 16, 95% CI 2-sided [12 to 21]
Statistical Analysis 8: Comparison: Group 3B vs Group B_0_1; Post booster/Post first dose-Adjusted geometric mean titers for 5/99 indicator strain were obtained by exponentiating (base 10) the least square means and the lower and upper limits of the 95% confidence intervals of the log-transformed titers obtained from an ANOVA estimation adjusting for vaccine group and country; Test type: Other — Vaccine comparison Post-booster or post-1st dose in V72_75 (Group 3B vs. Group B _0_1); ANOVA; Ratio of GMTs = 68, 95% CI 2-sided [51 to 90]
Statistical Analysis 9: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 15, analysis 7]; Test type: Other — Vaccine comparison- Pre-booster or pre-1st dose in V72_75 [Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; ANOVA; Ratio of GMTs = 18, 95% CI 2-sided [13 to 26]
Statistical Analysis 10: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 15, analysis 8]; Test type: Other — Vaccine comparison- post-booster or post-1st dose in V72_75 [Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; ANOVA; Ratio of GMTs = 74, 95% CI 2-sided [51 to 107]
Statistical Analysis 11: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 15, analysis 7]; Test type: Other — Vaccine comparison- Pre-booster or pre-1st dose in V72_75 [Group 3B (V72P10) vs. Group B_0_1 (V72P10)]; ANOVA; Ratio of GMTs = 14, 95% CI 2-sided [8.99 to 22]
Statistical Analysis 12: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 15, analysis 8]; Test type: Other — Vaccine comparison- post-booster or post-1st dose in V72_75 [Group 3B (V72P10) vs. Group B_0_1 (V72P10)]; ANOVA; Ratio of GMTs = 63, 95% CI 2-sided [41 to 95]
Statistical Analysis 13: Comparison: Group 3B vs Group B_0_1; Pre booster/Pre first dose-Adjusted geometric mean titers for NZ98/254 indicator strain were obtained by exponentiating (base 10) the least square means and the lower and upper limits of the 95% confidence intervals of the log-transformed titers obtained from an ANOVA estimation adjusting for vaccine group and country; Test type: Other — Vaccine comparison Pre-booster or pre-1st dose in V72_75 (Group 3B vs. Group B _0_1); ANOVA; Ratio of GMTs = 1.48, 95% CI 2-sided [1.24 to 1.75]
Statistical Analysis 14: Comparison: Group 3B vs Group B_0_1; Post booster dose/ post first dose-Adjusted geometric mean titers for NZ98/254 indicator strain were obtained by exponentiating (base 10) the least square means and the lower and upper limits of the 95% confidence intervals of the log-transformed titers obtained from an ANOVA estimation adjusting for vaccine group and country; Test type: Other — Vaccine comparison Post-booster or post-1st dose in V72_75 (Group 3B vs. Group B _0_1); ANOVA; Ratio of GMTs = 5.90, 95% CI 2-sided [4.49 to 7.76]
Statistical Analysis 15: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 15, analysis 13]; Test type: Other — Vaccine comparison- Pre-booster or pre-1st dose in V72_75 [Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; ANOVA; Ratio of GMTs = 1.32, 95% CI 2-sided [1.13 to 1.54]
Statistical Analysis 16: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); Post booster/Post first dose-Adjusted geometric mean titers for NZ98/254 indicator strain were obtained by exponentiating (base 10) the least square means and the lower and upper limits of the 95% confidence intervals of the log-transformed titers obtained from an ANOVA estimation adjusting for vaccine group and country; Test type: Other — Vaccine comparison- post-booster or post-1st dose in V72_75 [Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; ANOVA; Ratio of GMTs = 8.27, 95% CI 2-sided [5.83 to 12]
Statistical Analysis 17: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 15, analysis 13]; Test type: Other — Vaccine comparison- Pre-booster or pre-1st dose in V72_75 [Group 3B (V72P10) vs. Group B_0_1 (V72P10)]; ANOVA; Ratio of GMTs = 1.64, 95% CI 2-sided [1.22 to 2.20]
Statistical Analysis 18: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 15, analysis 16]; Test type: Other — Vaccine comparison- post-booster or post-1st dose in V72_75 [Group 3B (V72P10) vs. Group B_0_1 (V72P10)]; ANOVA; Ratio of GMTs = 4.36, 95% CI 2-sided [2.88 to 6.58]
Statistical Analysis 19: Comparison: Group 3B vs Group B_0_1; Pre booster/Pre first dose-Adjusted geometric mean titers for M10713 indicator strain were obtained by exponentiating (base 10) the least square means and the lower and upper limits of the 95% confidence intervals of the log-transformed titers obtained from an ANOVA estimation adjusting for vaccine group and country; Test type: Other — Vaccine comparison Pre-booster or pre-1st dose in V72_75 (Group 3B vs. Group B _0_1); ANOVA; Ratio of GMTs = 1.30, 95% CI 2-sided [0.97 to 1.75]
Statistical Analysis 20: Comparison: Group 3B vs Group B_0_1; Post booster/Post first dose-Adjusted geometric mean titers for M10713 indicator strain were obtained by exponentiating (base 10) the least square means and the lower and upper limits of the 95% confidence intervals of the log-transformed titers obtained from an ANOVA estimation adjusting for vaccine group and country; Test type: Other — Vaccine comparison Post-booster or post-1st dose in V72_75 (Group 3B vs. Group B _0_1); ANOVA; Ratio of GMTs = 2.60, 95% CI 2-sided [2.08 to 3.25]
Statistical Analysis 21: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 15, analysis 19]; Test type: Other — Vaccine comparison- Pre-booster or pre-1st dose in V72_75 [Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; ANOVA; Ratio of GMTs = 1.40, 95% CI 2-sided [0.90 to 2.18]
Statistical Analysis 22: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 15, analysis 20]; Test type: Other — Vaccine comparison- post-booster or post-1st dose in V72_75 [Group 3B (V72_41) vs. Group B_0_1 (V72_41)]; ANOVA; Ratio of GMTs = 2.79, 95% CI 2-sided [2.04 to 3.81]
Statistical Analysis 23: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 15, analysis 19]; Test type: Other — Vaccine comparison- Pre-booster or pre-1st dose in V72_75 [Group 3B (V72P10) vs. Group B_0_1 (V72P10)]; ANOVA; Ratio of GMTs = 1.23, 95% CI 2-sided [0.82 to 1.82]
Statistical Analysis 24: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 15, analysis 20]; Test type: Other — Vaccine comparison- post-booster or post-1st dose in V72_75 [Group 3B (V72P10) vs. Group B_0_1 (V72P10)]; ANOVA; Ratio of GMTs = 2.45, 95% CI 2-sided [1.79 to 3.36]

16. Secondary Outcome: Geometric Mean Ratio (GMRs) of GMTs After Booster Dose/First rMenB+OMV NZ Vaccination Versus Day 1.
Description: Bactericidal activity was measured against each of the fout N. meningitidis group B indicator strains H44/76,5/99,NZ98/254 and M10713 by calculating the GMRs of GMTs one month post-vaccination of a booster dose versus pre-booster dose (follow-on subjects) or first dose of rMenB+OMV NZ versus prefirst dose (naïve subjects) to each N. meningitidis group B indicator strain.
Time Frame: At Day 31 (30 days post booster dose/first dose of vaccination) versus Day 1 (prior to booster dose/first dose of vaccination).
Population: as for outcome 11
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Group 3B (V72_41) | Group 3B (V72P10) | Group 3B | Group B_0_1 (V72_41) | Group B_0_1 (V72P10) | Group B_0_1
Number analyzed (Participants) | 142 | 127 | 268 | 104 | 149 | 253
Ratio
  H44/76: number analyzed (Participants) | 141 | 127 | 268 | 104 | 149 | 253
  H44/76 | 65 [49 to 85] | 58 [44 to 76] | 61 [50 to 74] | 12 [8.69 to 16] | 16 [12 to 20] | 14 [11 to 17]
  5/99: number analyzed (Participants) | 118 | 93 | 211 | 96 | 129 | 225
  5/99 | 100 [72 to 139] | 64 [44 to 93] | 87 [67 to 112] | 25 [18 to 36] | 14 [9.90 to 19] | 20 [16 to 26]
  NZ98/254: number analyzed (Participants) | 142 | 118 | 260 | 103 | 146 | 249
  NZ98/254 | 23 [18 to 29] | 16 [12 to 22] | 19 [16 to 24] | 3.60 [2.69 to 4.81] | 6.43 [4.95 to 8.34] | 4.92 [3.97 to 6.10]
  M10713: number analyzed (Participants) | 140 | 127 | 267 | 103 | 149 | 252
  M10713 | 4.69 [3.72 to 5.92] | 5.16 [4.14 to 6.42] | 4.85 [4.10 to 5.72] | 2.37 [1.81 to 3.10] | 2.58 [2.11 to 3.16] | 2.44 [2.04 to 2.91]

17. Secondary Outcome: Percentages of Subjects With at Least 4-fold Increase in hSBA Titers Pre Vaccination Compared to One Month Post-booster/First rMenB+OMV NZ Vaccination
Description: The percentage of subjects with 4-fold rise at one month post-vaccination with a booster dose (follow-on subjects) /first dose (naive subjects) of rMenB+OMV NZ with respect to day 1 (follow-on subjects) / pre-first dose of rMenB+OMV NZ (naïve subjects). Percentage of subjects with four-fold rise in hSBA titers relative to baseline were defined as: • for a pre-vaccination titer < 4, a post-vaccination titer of at least 16; • for a pre-vaccination titer ≥ 4 but <LLOQ, a post vaccination titer of at least fourfold the LLOQ; • for a pre-vaccination titer ≥LLOQ, a post vaccination titer of at least fourfold the pre-vaccination titer
Time Frame: Group 3B: 1 month after booster dose; Group B_0_1: 1 month after first vaccination
Population: Analysis was performed on the Full Analysis set (FAS) booster. The FAS booster included all follow on subjects and all naive subjects in the All enrolled set who received vaccination at day 1 and provided evaluable immunogenicity result at day 31 for atleast one indicator strain.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Group 3B (V72_41) | Group 3B (V72P10) | Group 3B | Group B_0_1 (V72_41) | Group B_0_1 (V72P10) | Group B_0_1
Number analyzed (Participants) | 142 | 127 | 268 | 104 | 149 | 253
Percentage of subjects
  H44/76: number analyzed (Participants) | 141 | 127 | 268 | 104 | 149 | 253
  H44/76 | 95 [90.0 to 98.0] | 98 [93.3 to 99.51] | 96 [93.2 to 98.2] | 66 [56.4 to 75.3] | 72 [63.9 to 78.9] | 70 [63.5 to 75.2]
  5/99: number analyzed (Participants) | 118 | 93 | 211 | 96 | 129 | 225
  5/99 | 98 [94.0 to 99.79] | 97 [90.9 to 99.3] | 98 [94.6 to 99.2] | 79 [69.7 to 86.8] | 74 [65.2 to 81.0] | 76 [69.9 to 81.4]
  NZ98/254: number analyzed (Participants) | 142 | 118 | 260 | 103 | 146 | 249
  NZ98/254 | 83 [75.9 to 88.9] | 77 [68.5 to 84.3] | 80 [75.0 to 85.0] | 28 [19.7 to 37.9] | 53 [44.3 to 61.1] | 43 [36.3 to 49.0]
  M10713: number analyzed (Participants) | 140 | 127 | 267 | 103 | 149 | 252
  M10713 | 49 [40.0 to 57.2] | 49 [39.9 to 57.8] | 49 [42.6 to 54.9] | 24 [16.4 to 33.7] | 27 [19.9 to 34.7] | 26 [20.5 to 31.7]
Statistical Analysis 1: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 5, analysis 1]; Test type: Other — 1 month post booster/first dose of vaccination: Four-fold Increase (Group 3B vs. Group B_0_1) Difference; Miettinen and Nurminen score method; Vaccine group difference = 27, 95% CI 2-sided [20.7 to 33.0]
Statistical Analysis 2: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 5, analysis 1]; Test type: Other — 1 month post booster/first dose of vaccination: Four-fold Increase [Group 3B (V72_41) vs. Group B_0_1 (V72_41) Difference; Miettinen and Nurminen score method; Vaccine group difference = 29, 95% CI 2-sided [19.3 to 38.7]
Statistical Analysis 3: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 5, analysis 1]; Test type: Other — 1 month post booster/first dose of vaccination: Four-fold Increase [Group 3B (V72P10) vs. Group B_0_1 (V72P10) Difference; Miettinen and Nurminen score method; Vaccine group difference = 26, 95% CI 2-sided [18.3 to 33.9]
Statistical Analysis 4: Comparison: Group 3B vs Group B_0_1; The group difference in percentages of subjects with response against N. meningitidis serogroup B indicator strain 5/99 and the associated confidence interval or the difference was calculated using the method of Miettinen and Nurminen; Test type: Other — 1 month post booster/first dose of vaccination: Four-fold Increase (Group 3B vs. Group B_0_1) Difference; Miettinen and Nurminen score method; Vaccine group difference = 22, 95% CI 2-sided [15.9 to 27.9]
Statistical Analysis 5: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 5, analysis 4]; Test type: Other — [test comment as in outcome 17, analysis 2]; Miettinen and Nurminen score method; Vaccine group difference = 19, 95% CI 2-sided [11.5 to 28.5]
Statistical Analysis 6: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 5, analysis 4]; Test type: Other — [test comment as in outcome 17, analysis 3]; Miettinen and Nurminen score method; Vaccine group difference = 23, 95% CI 2-sided [14.6 to 31.9]
Statistical Analysis 7: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 5, analysis 7]; Test type: Other — 1 month post booster/first dose of vaccination: Four-fold Increase (Group 3B vs. Group B_0_1) Difference; Miettinen and Nurminen score method; Vaccine group difference = 38, 95% CI 2-sided [29.8 to 45.4]
Statistical Analysis 8: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 5, analysis 7]; Test type: Other — [test comment as in outcome 17, analysis 2]; Miettinen and Nurminen score method; Vaccine group difference = 55, 95% CI 2-sided [43.5 to 64.7]
Statistical Analysis 9: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 5, analysis 7]; Test type: Other — [test comment as in outcome 17, analysis 3]; Miettinen and Nurminen score method; Vaccine group difference = 24, 95% CI 2-sided [12.9 to 35.1]
Statistical Analysis 10: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 5, analysis 10]; Test type: Other — 1 month post booster/first dose of vaccination: Four-fold Increase (Group 3B vs. Group B_0_1) Difference; Miettinen and Nurminen score method; Vaccine group difference = 23, 95% CI 2-sided [14.7 to 30.8]
Statistical Analysis 11: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 5, analysis 10]; Test type: Other — [test comment as in outcome 17, analysis 2]; Miettinen and Nurminen score method; Vaccine group difference = 24, 95% CI 2-sided [12.2 to 35.5]
Statistical Analysis 12: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 5, analysis 10]; Test type: Other — [test comment as in outcome 17, analysis 3]; Miettinen and Nurminen score method; Vaccine group difference = 22, 95% CI 2-sided [10.6 to 32.9]

18. Secondary Outcome: Percentage of Subjects With hSBA ≥1:4 After Booster Dose/Second Vaccination of rMenB+OMV NZ
Description: Bactericidal activity was measured against the N. meningitidis group B indicator strains 5/99 and NZ98/254. On day 1, subjects in the Group B_0_1 were to be randomized into 2 different blood draw schedules according to a 1:1 ratio : 2 blood samples at different time points:
  Group B_0_1_1: blood draws at 3 and 30 days after the second dose. Group B_0_1_2: blood draws at 7 and 30 days after the second dose.
  This outcome measure was assessed only for strains 5/99 and NZ98/254.
Time Frame: Group 3B: 3, 7 and 30 days after third dose booster; Group B_0_1: At 3 (group B_0_1_1 only), 7 (sub-group B_0_1_2 only) and 30 days post-second dose.
Population: Analysis was performed on PPS kinetics which included all subjects who correctly received the vaccination at day 1/ day 1 & day 31 (naive subjects) & provided evaluable immunogenicity result at all of days 4, 8 & 31 (for follow-on subjects) or at all of days 34,38 and 61 (naive subjects).
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Group 3B (V72_41) | Group 3B (V72P10) | Group 3B | Group B_0_1 (V72_41) | Group B_0_1 (V72P10) | Group B_0_1
Number analyzed (Participants) | 130 | 103 | 233 | 94 | 109 | 203
Percentage of subjects
  5/99- 3 days post vaccination: number analyzed (Participants) | 103 | 82 | 185 | 44 | 42 | 86
  5/99- 3 days post vaccination | 78 [68.4 to 85.3] | 80 [70.3 to 88.4] | 79 [72.3 to 84.6] | 82 [67.3 to 91.8] | 88 [74.4 to 96.0] | 85 [75.5 to 91.7]
  5/99- 7 days post vaccination: number analyzed (Participants) | 103 | 82 | 185 | 40 | 48 | 88
  5/99- 7 days post vaccination | 100 [96.5 to 100.0] | 100 [95.6 to 100.0] | 100 [98.0 to 100.0] | 100 [91.2 to 100.0] | 98 [88.9 to 99.95] | 99 [93.8 to 99.97]
  5/99- 1 month post vaccination: number analyzed (Participants) | 103 | 82 | 185 | 84 | 90 | 174
  5/99- 1 month post vaccination | 100 [96.5 to 100.0] | 100 [95.6 to 100.0] | 100 [98.0 to 100.0] | 100 [95.7 to 100.0] | 98 [92.2 to 99.73] | 99 [95.9 to 99.86]
  NZ98/254- 3 days post vaccination: number analyzed (Participants) | 130 | 103 | 233 | 50 | 55 | 105
  NZ98/254- 3 days post vaccination | 12 [6.6 to 18.3] | 28 [19.7 to 37.9] | 19 [14.1 to 24.5] | 32 [19.5 to 46.7] | 60 [45.9 to 73.0] | 47 [36.9 to 56.7]
  NZ98/254- 7 days post vaccination: number analyzed (Participants) | 130 | 103 | 233 | 44 | 54 | 98
  NZ98/254- 7 days post vaccination | 73 [64.6 to 80.5] | 80 [70.5 to 86.9] | 76 [70.0 to 81.3] | 80 [64.7 to 90.2] | 81 [68.6 to 90.7] | 81 [71.4 to 87.9]
  NZ98/254- 1 month post vaccination | 94 [88.2 to 97.3] | 94 [87.8 to 97.8] | 94 [90.1 to 96.7] | 82 [72.6 to 89.1] | 79 [70.0 to 86.1] | 80 [74.1 to 85.5]
Statistical Analysis 1: Comparison: Group 3B vs Group B_0_1; 3 days post vaccination-The group difference in percentages of subjects with response against N. meningitidis serogroup B indicator strain 5/99 and the associated confidence interval for the difference was calculated using the method of Miettinen and Nurminen; Test type: Other — Vaccine comparison at Day 4 Group 3B vs Day 34 Group B_0_1 (3 days after booster or 2nd dose); Miettinen and Nurminen score method — Vaccine comparison at Day 4 Group 3B vs Day 34 Group B_0_1 (3 days after booster or 2nd dose); Vaccine group difference = -6, 95% CI 2-sided [-15.0 to 4.5]
Statistical Analysis 2: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 18, analysis 1]; Test type: Other — Vaccine comparison at Day 4 Group 3B (V72_41) vs Day 34 Group B_0_1 (V72_41) (3 days after booster or 2nd dose); Miettinen and Nurminen score method; Vaccine group difference = -4, 95% CI 2-sided [-17.0 to 11.4]
Statistical Analysis 3: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 18, analysis 1]; Test type: Other — Vaccine comparison at Day 4 Group 3B (V72P10) vs Day 34 Group B_0_1 (V72P10) (3 days after booster or 2nd dose); Miettinen and Nurminen score method; Vaccine group difference = -8, 95% CI 2-sided [-20.0 to 7.3]
Statistical Analysis 4: Comparison: Group 3B vs Group B_0_1; 7 days post vaccination-The group difference in percentages of subjects with response against N. meningitidis serogroup B indicator strain 5/99 and the associated confidence interval for the difference was calculated using the method of Miettinen and Nurminen; Test type: Other — Vaccine comparison at Day 8 Group 3B vs Day 38 Group B_0_1 (7 days after booster or 2nd dose); Miettinen and Nurminen score method; Vaccine group difference = 1, 95% CI 2-sided [-0.9 to 6.2]
Statistical Analysis 5: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 18, analysis 4]; Test type: Other — Vaccine comparison at Day 8 Group 3B (V72_41) vs Day 38 Group B_0_1 (V72_41) (7 days after booster or 2nd dose); Miettinen and Nurminen score method; Vaccine group difference = 0, 95% CI 2-sided [-3.6 to 8.8]
Statistical Analysis 6: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 18, analysis 4]; Test type: Other — Vaccine comparison at Day 8 Group 3B (V72P10) vs Day 34 Group B_0_1 (V72P10) (7 days after booster or 2nd dose); Miettinen and Nurminen score method; Vaccine group difference = 2, 95% CI 2-sided [-2.5 to 11.0]
Statistical Analysis 7: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); 1 month post vaccination-The group difference in percentages of subjects with response against N. meningitidis serogroup B indicator strain 5/99 and the associated confidence interval for the difference was calculated using the method of Miettinen and Nurminen; Test type: Other — Vaccine comparison at Day 31 Group 3B (V72_41) vs Day 61 Group B_0_1(V72_41) (1 month after booster or 2nd dose); Miettinen and Nurminen score method; Vaccine group difference = 0, 95% CI 2-sided [-3.6 to 4.4]
Statistical Analysis 8: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 18, analysis 7]; Test type: Other — Vaccine comparison at Day 31 Group 3B (V72P10) vs Day 61 Group B_0_1 (V72P10) (1 month after booster or 2nd dose); Miettinen and Nurminen score method; Vaccine group difference = 2, 95% CI 2-sided [-2.3 to 7.8]
Statistical Analysis 9: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 18, analysis 7]; Test type: Other — Vaccine comparison at Day 31 Group 3B vs Day 61 Group B_0_1 (1 month after booster or 2nd dose); Miettinen and Nurminen score method; Vaccine group difference = 1, 95% CI 2-sided [-0.9 to 4.1]
Statistical Analysis 10: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); 3 days post vaccination-The group difference in percentages of subjects with response against N. meningitidis serogroup B indicator strain NZ98/254 and the associated confidence interval for the difference was calculated using the method of Miettinen and Nurminen; Test type: Other — Vaccine comparison at Day 4 Group 3B (V72_41) vs Day 34 Group B_0_1 (V72_41) (3 days after booster or 2nd dose); Miettinen and Nurminen score method; Vaccine group difference = -20, 95% CI 2-sided [-35.2 to -7.5]
Statistical Analysis 11: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 18, analysis 10]; Test type: Other — Vaccine comparison at Day 4 Group 3B (V72P10) vs Day 34 Group B_0_1 (V72P10) (3 days after booster or 2nd dose); Miettinen and Nurminen score method; Vaccine group difference = -32, 95% CI 2-sided [-46.5 to -15.7]
Statistical Analysis 12: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 18, analysis 10]; Test type: Other — Vaccine comparison at Day 4 Group 3B vs Day 34 Group B_0_1 (3 days after booster or 2nd dose); Miettinen and Nurminen score method; Vaccine group difference = -28, 95% CI 2-sided [-38.4 to -17.1]
Statistical Analysis 13: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); 7 days post vaccination-The group difference in percentages of subjects with response against N. meningitidis serogroup B indicator strain NZ98/254 and the associated confidence interval for the difference was calculated using the method of Miettinen and Nurminen; Test type: Other — Vaccine comparison at Day 8 Group 3B (V72_41) vs Day 38 Group B_0_1 (V72_41) (7 days after booster or 2nd dose); Miettinen and Nurminen score method; Vaccine group difference = -6, 95% CI 2-sided [-19.2 to 9.2]
Statistical Analysis 14: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 18, analysis 13]; Test type: Other — Vaccine comparison at Day 8 Group 3B (V72_41) vs Day 38 Group B_0_1 (V72_41) (7 days after booster or 2nd dose); Miettinen and Nurminen score method; Vaccine group difference = -2, 95% CI 2-sided [-14.1 to 12.3]
Statistical Analysis 15: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 18, analysis 13]; Test type: Other — Vaccine comparison at Day 8 Group 3B vs Day 38 Group B_0_1 (7 days after booster or 2nd dose); Miettinen and Nurminen score method; Vaccine group difference = -5, 95% CI 2-sided [-13.6 to 5.6]
Statistical Analysis 16: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); 1 month post vaccination-The group difference in percentages of subjects with response against N. meningitidis serogroup B indicator strain NZ98/254 and the associated confidence interval for the difference was calculated using the method of Miettinen and Nurminen; Test type: Other — Vaccine comparison at Day 31 Group 3B (V72_41) vs Day 61 Group B_0_1 (V72_41) (1 month after booster or 2nd dose); Miettinen and Nurminen score method; Vaccine group difference = 12, 95% CI 2-sided [3.6 to 21.6]
Statistical Analysis 17: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 18, analysis 16]; Test type: Other — Vaccine comparison at Day 31 Group 3B (V72P10) vs Day 61 Group B_0_1 (V72P10) (1 month after booster or 2nd dose); Miettinen and Nurminen score method; Vaccine group difference = 15, 95% CI 2-sided [6.4 to 24.6]
Statistical Analysis 18: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 18, analysis 16]; Test type: Other — Vaccine comparison at Day 31 Group 3B vs Day 61 Group B_0_1 (1 month after booster or 2nd dose); Miettinen and Nurminen score method; Vaccine group difference = 14, 95% CI 2-sided [7.6 to 20.3]

19. Secondary Outcome: Percentage of Subjects With hSBA ≥1:5 After Booster Dose/Second Vaccination of rMenB+OMV NZ
Description: Bactericidal activity was measured against the N. meningitidis group B indicator strains H44/76 and M10713. On day 1, subjects in the Group B_0_1 were to be randomized into 2 different blood draw schedules according to a 1:1 ratio : 2 blood samples at different time points:
  Group B_0_1_1: blood draws at 3 and 30 days after the second dose. Group B_0_1_2: blood draws at 7 and 30 days after the second dose. This outcome measure was assessed only for strains H44/76 and M10713.
Time Frame: Group 3B: 3, 7 and 30 days after third dose booster; Group B_0_1: At 3 (group B_0_1_1 only), 7 (sub-group B_0_1_2 only) and 30 days post-second dose."
Population: Analysis was performed on the PPS kinetics which included all subjects who correctly received the vaccination at day 1/ day 1 & day 31 (naive subjects) & provided evaluable immunogenicity result at all of days 4, 8 & 31 (for follow-on subjects) or at all of days 34,38 & 61 (naive subjects).
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Group 3B (V72_41) | Group 3B (V72P10) | Group 3B | Group B_0_1 (V72_41) | Group B_0_1 (V72P10) | Group B_0_1
Number analyzed (Participants) | 130 | 112 | 242 | 94 | 109 | 203
Percentage of subjects
  H44/76 3 days post vaccination: number analyzed (Participants) | 130 | 112 | 242 | 50 | 55 | 105
  H44/76 3 days post vaccination | 28 [20.9 to 37.0] | 46 [36.1 to 55.2] | 36 [30.3 to 42.8] | 74 [59.7 to 85.4] | 85 [73.3 to 93.5] | 80 [71.1 to 87.2]
  H44/76 7 days post vaccination: number analyzed (Participants) | 130 | 112 | 242 | 44 | 54 | 98
  H44/76 7 days post vaccination | 97 [92.3 to 99.2] | 99 [95.1 to 99.98] | 98 [95.2 to 99.3] | 100 [92.0 to 100.0] | 98 [90.1 to 99.95] | 99 [94.4 to 99.97]
  H44/76 1 month post vaccination | 98 [93.4 to 99.52] | 100 [96.8 to 100.0] | 99 [96.4 to 99.74] | 99 [94.2 to 99.97] | 99 [95.0 to 99.98] | 99 [96.5 to 99.88]
  M10713- 3 days post-vaccination: number analyzed (Participants) | 129 | 112 | 241 | 50 | 55 | 105
  M10713- 3 days post-vaccination | 71 [62.7 to 78.9] | 86 [77.8 to 91.6] | 78 [72.2 to 83.1] | 76 [61.8 to 86.9] | 87 [75.5 to 94.7] | 82 [73.2 to 88.7]
  M10713- 7 days post-vaccination: number analyzed (Participants) | 129 | 112 | 241 | 44 | 54 | 98
  M10713- 7 days post-vaccination | 98 [93.4 to 99.52] | 97 [92.4 to 99.4] | 98 [94.7 to 99.1] | 95 [84.5 to 99.4] | 96 [87.3 to 99.55] | 96 [89.9 to 98.9]
  M10713- 1 month post-vaccination: number analyzed (Participants) | 129 | 112 | 241 | 94 | 109 | 203
  M10713- 1 month post-vaccination | 99 [95.8 to 99.98] | 99 [95.1 to 99.98] | 99 [97.0 to 99.90] | 90 [82.6 to 95.5] | 95 [89.6 to 98.5] | 93 [88.7 to 96.2]
Statistical Analysis 1: Comparison: Group 3B vs Group B_0_1; 3 days post vaccination-The group difference in percentages of subjects with response against N. meningitidis serogroup B indicator strain H44/76 and the associated confidence interval for the difference was calculated using the method of Miettinen and Nurminen; Test type: Other — Vaccine comparison at Day 4 Group 3B vs Day 34 Group B_0_1 (3 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -44, 95% CI 2-sided [-52.7 to -33.1]
Statistical Analysis 2: Comparison: Group 3B vs Group B_0_1; 7 days post vaccination-The group difference in percentages of subjects with response against N. meningitidis serogroup B indicator strain H44/76 and the associated confidence interval for the difference was calculated using the method of Miettinen and Nurminen; Test type: Other — Vaccine comparison at Day 8 Group 3B vs Day 38 Group B_0_1 (7 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -1, 95% CI 2-sided [-3.9 to 3.6]
Statistical Analysis 3: Comparison: Group 3B vs Group B_0_1; 1 month post vaccination-The group difference in percentages of subjects with response against N. meningitidis serogroup B indicator strain H44/76 and the associated confidence interval for the difference was calculated using the method of Miettinen and Nurminen; Test type: Other — Vaccine comparison at Day 31 Group 3B vs Day 61 Group B_0_1 (1 month after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 0, 95% CI 2-sided [-2.7 to 2.4]
Statistical Analysis 4: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 19, analysis 1]; Test type: Other — Vaccine comparison at Day 4 Group 3B (V72_41) vs Day 34 Group B_0_1 (V72_41) (3 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -46, 95% CI 2-sided [-58.4 to -29.8]
Statistical Analysis 5: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 19, analysis 2]; Test type: Other — Vaccine comparison at Day 8 Group 3B (V72_41) vs Day 38 Group B_0_1 (V72_41) (7 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -3, 95% CI 2-sided [-7.7 to 5.1]
Statistical Analysis 6: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 19, analysis 3]; Test type: Other — Vaccine comparison at Day 31 Group 3B (V72_41) vs Day 61 Group B_0_1 (V72_41) (1 month after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -1, 95% CI 2-sided [-5.7 to 3.7]
Statistical Analysis 7: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 19, analysis 1]; Test type: Other — Vaccine comparison at Day 4 Group 3B (V72P10) vs Day 34 Group B_0_1 (V72P10) (3 days after booster or 2nd dose); Miettinen and Nurminen score method; Vaccine group difference = -40, 95% CI 2-sided [-51.8 to -25.4]
Statistical Analysis 8: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 19, analysis 2]; Test type: Other — Vaccine comparison at Day 8 Group 3B (V72P10) vs Day 38 Group B_0_1 (V72P10) (7 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 1, 95% CI 2-sided [-3.3 to 9.0]
Statistical Analysis 9: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 19, analysis 3]; Test type: Other — Vaccine comparison at Day 31 Group 3B (V72P10) vs Day 61 Group B_0_1 (V72P10) (1 month after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 1, 95% CI 2-sided [-2.4 to 5.0]
Statistical Analysis 10: Comparison: Group 3B vs Group B_0_1; 3 days post vaccination-The group difference in percentages of subjects with response N. meningitidis serogroup B indicator strain M10713 and the associated confidence interval for the difference was calculated using the method of Miettinen and Nurminen; Test type: Other — Vaccine comparison at Day 4 Group 3B vs Day 34 Group B_0_1 (3 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -4, 95% CI 2-sided [-12.4 to 5.8]
Statistical Analysis 11: Comparison: Group 3B vs Group B_0_1; 7 days post vaccination-The group difference in percentages of subjects with response N. meningitidis serogroup B indicator strain M10713 and the associated confidence interval for the difference was calculated using the method of Miettinen and Nurminen; Test type: Other — Vaccine comparison at Day 8 Group 3B vs Day 38 Group B_0_1 (7 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 2, 95% CI 2-sided [-2.2 to 7.7]
Statistical Analysis 12: Comparison: Group 3B vs Group B_0_1; 1 month post vaccination-The group difference in percentages of subjects with response N. meningitidis serogroup B indicator strain M10713 and the associated confidence interval for the difference was calculated using the method of Miettinen and Nurminen; Test type: Other — Vaccine comparison at Day 31 Group 3B vs Day 61 Group B_0_1 (1 month after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 6, 95% CI 2-sided [2.8 to 10.5]
Statistical Analysis 13: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); 3 days post vaccination-The group difference in percentages of subjects with response against N. meningitidis serogroup B indicator strain M10713 and the associated confidence interval for the difference was calculated using the method of Miettinen and Nurminen; Test type: Other — Vaccine comparison at Day 4 Group 3B (V72_41) vs Day 34 Group B_0_1 (V72_41) (3 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -5, 95% CI 2-sided [-17.8 to 10.6]
Statistical Analysis 14: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); 7 days post vaccination-The group difference in percentages of subjects with response against N. meningitidis serogroup B indicator strain M10713 and the associated confidence interval for the difference was calculated using the method of Miettinen and Nurminen; Test type: Other — Vaccine comparison at Day 8 Group 3B (V72_41) vs Day 38 Group B_0_1 (V72_41) (7 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 2, 95% CI 2-sided [-3.2 to 13.0]
Statistical Analysis 15: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); 1 month post vaccination-The group difference in percentages of subjects with response against N. meningitidis serogroup B indicator strain M10713 and the associated confidence interval for the difference was calculated using the method of Miettinen and Nurminen; Test type: Other — Vaccine comparison at Day 31 Group 3B (V72_41) vs Day 61 Group B_0_1 (V72_41) (1 month after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 9, 95% CI 2-sided [3.7 to 16.5]
Statistical Analysis 16: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 19, analysis 13]; Test type: Other — Vaccine comparison at Day 4 Group 3B (V72P10) vs Day 34 Group B_0_1 (V72P10) (3 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -2, 95% CI 2-sided [-11.8 to 11.0]
Statistical Analysis 17: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 19, analysis 14]; Test type: Other — Vaccine comparison at Day 8 Group 3B (V72_41) vs Day 38 Group B_0_1 (V72_41) (7 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 1, 95% CI 2-sided [-4.6 to 10.1]
Statistical Analysis 18: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 19, analysis 15]; Test type: Other — Vaccine comparison at Day 31 Group 3B (V72P10) vs Day 61 Group B_0_1 (V72P10) (1 month days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 4, 95% CI 2-sided [-0.8 to 9.5]

20. Secondary Outcome: Percentage of Subjects With hSBA ≥1:8 After Booster Dose/Second Vaccination of rMenB+OMV NZ
Description: Bactericidal activity was measured against each of the four N. meningitidis group B indicator strains H44/76,5/99,NZ98/254 and M10713. On day 1, subjects in the Group B_0_1 were to be randomized into 2 different blood draw schedules according to a 1:1 ratio : 2 blood samples at different time points:
  Group B_0_1_1: blood draws at 3 and 30 days after the second dose. Group B_0_1_2: blood draws at 7 and 30 days after the second dose.
Time Frame: as for outcome 18
Population: Analysis was performed on PPS kinetics which included all subjects who had no protocol deviations/any other reason defined prior to analysis, leading to exclusion & correctly received the vaccination at day 1/day 31 & day 1 & provided evaluable immunogenicity result at all of days 4, 8 & 31 (follow-on subjects)or at all of days 34, 38 & 61(naive)
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Group 3B (V72_41) | Group 3B (V72P10) | Group 3B | Group B_0_1 (V72_41) | Group B_0_1 (V72P10) | Group B_0_1
Number analyzed (Participants) | 130 | 112 | 242 | 94 | 109 | 203
Percentage of subjects
  H44/76 3 days post vaccination: number analyzed (Participants) | 130 | 112 | 242 | 50 | 55 | 105
  H44/76 3 days post vaccination | 22 [15.5 to 30.4] | 39 [30.2 to 49.0] | 30 [24.5 to 36.4] | 70 [55.4 to 82.1] | 80 [67.0 to 89.6] | 75 [65.9 to 83.1]
  H44/76 7 days post vaccination: number analyzed (Participants) | 130 | 112 | 242 | 44 | 54 | 98
  H44/76 7 days post vaccination | 95 [89.2 to 97.8] | 98 [93.7 to 99.78] | 96 [93.1 to 98.3] | 95 [84.5 to 99.4] | 98 [90.1 to 99.95] | 97 [91.3 to 99.4]
  H44/76 1 month post vaccination | 98 [93.4 to 99.52] | 100 [96.8 to 100.0] | 99 [96.4 to 99.74] | 99 [94.2 to 99.97] | 97 [92.2 to 99.4] | 98 [95.0 to 99.5]
  5/99- 3 days post-vaccination: number analyzed (Participants) | 103 | 82 | 185 | 44 | 42 | 86
  5/99- 3 days post-vaccination | 74 [64.2 to 82.0] | 79 [68.9 to 87.4] | 76 [69.4 to 82.2] | 80 [64.7 to 90.2] | 86 [71.5 to 94.6] | 83 [72.9 to 89.9]
  5/99- 7 days post-vaccination: number analyzed (Participants) | 103 | 82 | 185 | 40 | 48 | 88
  5/99- 7 days post-vaccination | 100 [96.5 to 100.0] | 100 [95.6 to 100.0] | 100 [98.0 to 100.0] | 100 [91.2 to 100.0] | 98 [88.9 to 99.95] | 99 [93.8 to 99.97]
  5/99- 1 month post-vaccination: number analyzed (Participants) | 103 | 82 | 185 | 84 | 90 | 174
  5/99- 1 month post-vaccination | 100 [96.5 to 100.0] | 100 [95.6 to 100.0] | 100 [98.0 to 100.0] | 100 [95.7 to 100.0] | 98 [92.2 to 99.73] | 99 [95.9 to 99.86]
  NZ98/254- 3 days post-vaccination: number analyzed (Participants) | 130 | 103 | 233 | 50 | 55 | 105
  NZ98/254- 3 days post-vaccination | 10 [5.4 to 16.5] | 23 [15.5 to 32.7] | 16 [11.4 to 21.2] | 28 [16.2 to 42.5] | 55 [40.6 to 68.0] | 42 [32.3 to 51.9]
  NZ98/254- 7 days post-vaccination: number analyzed (Participants) | 130 | 103 | 233 | 44 | 54 | 98
  NZ98/254- 7 days post-vaccination | 61 [51.8 to 69.2] | 74 [64.2 to 82.0] | 67 [60.1 to 72.6] | 68 [52.4 to 81.4] | 70 [56.4 to 82.0] | 69 [59.3 to 78.3]
  NZ98/254- 1 month post-vaccination: number analyzed (Participants) | 130 | 103 | 233 | 94 | 109 | 203
  NZ98/254- 1 month post-vaccination | 85 [77.2 to 90.3] | 91 [84.1 to 95.9] | 88 [82.6 to 91.5] | 65 [54.4 to 74.5] | 69 [59.2 to 77.3] | 67 [60.1 to 73.4]
  M10713- 3 days post-vaccination: number analyzed (Participants) | 129 | 112 | 241 | 50 | 55 | 105
  M10713- 3 days post-vaccination | 62 [53.1 to 70.4] | 79 [69.8 to 85.8] | 70 [63.5 to 75.4] | 62 [47.2 to 75.3] | 84 [71.2 to 92.2] | 73 [63.8 to 81.5]
  M10713- 7 days post-vaccination: number analyzed (Participants) | 129 | 112 | 241 | 44 | 54 | 98
  M10713- 7 days post-vaccination | 95 [90.2 to 98.3] | 96 [89.9 to 98.5] | 95 [92.0 to 97.7] | 93 [81.3 to 98.6] | 94 [84.6 to 98.8] | 94 [87.1 to 97.7]
  M10713- 1 month post-vaccination: number analyzed (Participants) | 129 | 112 | 241 | 94 | 109 | 203
  M10713- 1 month post-vaccination | 98 [94.5 to 99.81] | 98 [93.7 to 99.78] | 98 [95.8 to 99.55] | 86 [77.5 to 92.4] | 94 [87.2 to 97.4] | 90 [85.2 to 93.9]
Statistical Analysis 1: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 19, analysis 1]; Test type: Other — Vaccine comparison at Day 4 Group 3B vs Day 34 Group B_0_1 (3 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -45, 95% CI 2-sided [-54.4 to -34.3]
Statistical Analysis 2: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 19, analysis 2]; Test type: Other — Vaccine comparison at Day 8 Group 3B vs Day 38 Group B_0_1 (7 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -1, 95% CI 2-sided [-4.5 to 5.2]
Statistical Analysis 3: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 19, analysis 3]; Test type: Other — Vaccine comparison at Day 31 Group 3B vs Day 61 Group B_0_1 (1 month after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 1, 95% CI 2-sided [-1.9 to 3.9]
Statistical Analysis 4: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 19, analysis 1]; Test type: Other — Vaccine comparison at Day 4 Group 3B (V72_41) vs Day 34 Group B_0_1 (V72_41) (3 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -48, 95% CI 2-sided [-60.8 to -32.0]
Statistical Analysis 5: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 19, analysis 2]; Test type: Other — Vaccine comparison at Day 8 Group 3B (V72_41) vs Day 38 Group B_0_1 (V72_41) (7 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -1, 95% CI 2-sided [-7.3 to 10.1]
Statistical Analysis 6: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 19, analysis 3]; Test type: Other — Vaccine comparison at Day 31 Group 3B (V72_41) vs Day 61 Group B_0_1 (V72_41) (1 month after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -1, 95% CI 2-sided [-5.7 to 3.7]
Statistical Analysis 7: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 19, analysis 1]; Test type: Other — Vaccine comparison at Day 4 Group 3B (V72P10) vs Day 34 Group B_0_1 (V72P10) (3 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -41, 95% CI 2-sided [-53.3 to -25.5]
Statistical Analysis 8: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 19, analysis 2]; Test type: Other — Vaccine comparison at Day 8 Group 3B (V72P10) vs Day 38 Group B_0_1 (V72P10) (7 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 0, 95% CI 2-sided [-4.8 to 8.1]
Statistical Analysis 9: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 19, analysis 3]; Test type: Other — Vaccine comparison at Day 31 Group 3B (V72P10) vs Day 61 Group B_0_1 (V72P10) (1 month days after booster or 2nd dose); Miettinen and Nurminen score methodx; vaccine group difference = 3, 95% CI 2-sided [-0.6 to 7.8]
Statistical Analysis 10: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 18, analysis 1]; Test type: Other — Vaccine comparison at Day 4 Group 3B vs Day 34 Group B_0_1 (3 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -6, 95% CI 2-sided [-15.9 to 4.6]
Statistical Analysis 11: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 18, analysis 4]; Test type: Other — Vaccine comparison at Day 8 Group 3B vs Day 38 Group B_0_1 (7 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 1, 95% CI 2-sided [-0.9 to 6.2]
Statistical Analysis 12: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 18, analysis 7]; Test type: Other — Vaccine comparison at Day 31 Group 3B vs Day 61 Group B_0_1 (1 month after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 1, 95% CI 2-sided [-0.9 to 4.1]
Statistical Analysis 13: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 18, analysis 1]; Test type: Other — Vaccine comparison at Day 4 Group 3B (V72_41) vs Day 34 Group B_0_1 (V72_41) (3 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -6, 95% CI 2-sided [-19.2 to 10.3]
Statistical Analysis 14: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 18, analysis 4]; Test type: Other — Vaccine comparison at Day 8 Group 3B (V72_41) vs Day 38 Group B_0_1 (V72_41) (7 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 0, 95% CI 2-sided [-3.6 to 8.8]
Statistical Analysis 15: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 18, analysis 7]; Test type: Other — Vaccine comparison at Day 31 Group 3B (V72_41) vs Day 61 Group B_0_1 (V72_41) (1 month after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 0, 95% CI 2-sided [-3.6 to 4.4]
Statistical Analysis 16: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 18, analysis 1]; Test type: Other — Vaccine comparison at Day 4 Group 3B (V72P10) vs Day 34 Group B_0_1 (V72P10) (3 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -6, 95% CI 2-sided [-19.4 to 9.1]
Statistical Analysis 17: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 18, analysis 4]; Test type: Other — Vaccine comparison at Day 8 Group 3B (V72P10) vs Day 38 Group B_0_1 (V72P10) (7 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 2, 95% CI 2-sided [-2.5 to 11.0]
Statistical Analysis 18: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 18, analysis 7]; Test type: Other — Vaccine comparison at Day 31 Group 3B (V72P10) vs Day 61 Group B_0_1 (V72P10) (1 month days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 2, 95% CI 2-sided [-2.3 to 7.8]
Statistical Analysis 19: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 18, analysis 10]; Test type: Other — Vaccine comparison at Day 4 Group 3B vs Day 34 Group B_0_1 (3 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -26, 95% CI 2-sided [-36.6 to -15.7]
Statistical Analysis 20: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 18, analysis 13]; Test type: Other — Vaccine comparison at Day 8 Group 3B vs Day 38 Group B_0_1 (7 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -3, 95% CI 2-sided [-13.3 to 8.5]
Statistical Analysis 21: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 18, analysis 16]; Test type: Other — Vaccine comparison at Day 31 Group 3B vs Day 61 Group B_0_1 (1 month after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 21, 95% CI 2-sided [12.8 to 28.3]
Statistical Analysis 22: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 18, analysis 10]; Test type: Other — Vaccine comparison at Day 4 Group 3B (V72_41) vs Day 34 Group B_0_1 (V72_41) (3 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -18, 95% CI 2-sided [-32.5 to -5.8]
Statistical Analysis 23: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 18, analysis 13]; Test type: Other — Vaccine comparison at Day 8 Group 3B (V72_41) vs Day 38 Group B_0_1 (V72_41) (7 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -7, 95% CI 2-sided [-22.3 to 9.5]
Statistical Analysis 24: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 18, analysis 16]; Test type: Other — Vaccine comparison at Day 31 Group 3B (V72_41) vs Day 61 Group B_0_1 (V72_41) (1 month after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 20, 95% CI 2-sided [8.4 to 31.3]
Statistical Analysis 25: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 18, analysis 10]; Test type: Other — Vaccine comparison at Day 4 Group 3B (V72P10) vs Day 34 Group B_0_1 (V72P10) (3 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -31, 95% CI 2-sided [-46.0 to -15.5]
Statistical Analysis 26: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 18, analysis 13]; Test type: Other — Vaccine comparison at Day 8 Group 3B (V72P10) vs Day 38 Group B_0_1 (V72P10) (7 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 3, 95% CI 2-sided [-10.8 to 18.8]
Statistical Analysis 27: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 18, analysis 16]; Test type: Other — Vaccine comparison at Day 31 Group 3B (V72P10) vs Day 61 Group B_0_1 (V72P10) (1 month days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 22, 95% CI 2-sided [12.1 to 32.8]
Statistical Analysis 28: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 19, analysis 13]; Test type: Other — Vaccine comparison at Day 4 Group 3B vs Day 34 Group B_0_1 (3 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -4, 95% CI 2-sided [-13.4 to 7.1]
Statistical Analysis 29: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 19, analysis 14]; Test type: Other — Vaccine comparison at Day 8 Group 3B vs Day 38 Group B_0_1 (7 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 2, 95% CI 2-sided [-3.2 to 8.5]
Statistical Analysis 30: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 19, analysis 15]; Test type: Other — Vaccine comparison at Day 31 Group 3B vs Day 61 Group B_0_1 (1 month after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 8, 95% CI 2-sided [4.2 to 13.2]
Statistical Analysis 31: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 19, analysis 13]; Test type: Other — Vaccine comparison at Day 4 Group 3B (V72_41) vs Day 34 Group B_0_1 (V72_41) (3 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 0, 95% CI 2-sided [-15.1 to 16.1]
Statistical Analysis 32: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 19, analysis 14]; Test type: Other — Vaccine comparison at Day 8 Group 3B (V72_41) vs Day 38 Group B_0_1 (V72_41) (7 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 2, 95% CI 2-sided [-4.7 to 13.9]
Statistical Analysis 33: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 19, analysis 15]; Test type: Other — Vaccine comparison at Day 31 Group 3B (V72_41) vs Day 61 Group B_0_1 (V72_41) (1 month after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 12, 95% CI 2-sided [5.9 to 20.9]
Statistical Analysis 34: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 19, analysis 13]; Test type: Other — Vaccine comparison at Day 4 Group 3B (V72P10) vs Day 34 Group B_0_1 (V72P10) (3 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -5, 95% CI 2-sided [-16.7 to 8.6]
Statistical Analysis 35: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 19, analysis 14]; Test type: Other — Vaccine comparison at Day 8 Group 3B (V72P10) vs Day 38 Group B_0_1 (V72P10) (7 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 1, 95% CI 2-sided [-5.7 to 11.1]
Statistical Analysis 36: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 19, analysis 15]; Test type: Other — Vaccine comparison at Day 31 Group 3B (V72P10) vs Day 61 Group B_0_1 (V72P10) (1 month after booster or 2nd dose); vaccine group difference = 5, 95% CI 2-sided [-0.7 to 11.1]

21. Secondary Outcome: Percentage of Subjects With hSBA ≥1:16 After Booster Dose/Second Vaccination of rMenB+OMV NZ
Description: as for outcome 20
Time Frame: as for outcome 18
Population: as for outcome 20
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Group 3B (V72_41) | Group 3B (V72P10) | Group 3B | Group B_0_1 (V72_41) | Group B_0_1 (V72P10) | Group B_0_1
Number analyzed (Participants) | 130 | 112 | 242 | 94 | 109 | 203
Percentage of subjects
  H44/76 3 days post vaccination: number analyzed (Participants) | 130 | 112 | 242 | 50 | 55 | 105
  H44/76 3 days post vaccination | 13 [7.8 to 20.1] | 29 [21.2 to 38.8] | 21 [15.7 to 26.3] | 40 [26.4 to 54.8] | 60 [45.9 to 73.0] | 50 [40.5 to 60.4]
  H44/76 7 days post vaccination: number analyzed (Participants) | 130 | 112 | 242 | 44 | 54 | 98
  H44/76 7 days post vaccination | 92 [85.4 to 95.7] | 98 [93.7 to 99.78] | 95 [91.0 to 97.1] | 89 [75.4 to 96.2] | 94 [84.6 to 98.8] | 92 [84.5 to 96.4]
  H44/76 1 month post vaccination | 98 [93.4 to 99.52] | 100 [96.8 to 100.0] | 99 [96.4 to 99.74] | 90 [82.6 to 95.5] | 92 [84.9 to 96.2] | 91 [86.3 to 94.7]
  5/99- 3 days post-vaccination: number analyzed (Participants) | 103 | 82 | 185 | 44 | 42 | 86
  5/99- 3 days post-vaccination | 69 [59.1 to 77.7] | 72 [60.9 to 81.3] | 70 [63.1 to 76.8] | 75 [59.7 to 86.8] | 76 [60.5 to 87.9] | 76 [65.1 to 84.2]
  5/99- 7 days post-vaccination: number analyzed (Participants) | 103 | 82 | 185 | 40 | 48 | 88
  5/99- 7 days post-vaccination | 100 [96.5 to 100] | 100 [95.6 to 100] | 100 [98.0 to 100.0] | 100 [91.2 to 100] | 98 [88.9 to 99.95] | 99 [93.8 to 99.97]
  5/99- 1 month post-vaccination: number analyzed (Participants) | 103 | 82 | 185 | 84 | 90 | 174
  5/99- 1 month post-vaccination | 100 [96.5 to 100.0] | 100 [95.6 to 100.0] | 100 [98.0 to 100.0] | 100 [95.7 to 100.0] | 97 [90.6 to 99.3] | 98 [95.0 to 99.64]
  NZ98/254- 3 days post-vaccination: number analyzed (Participants) | 130 | 103 | 233 | 50 | 55 | 105
  NZ98/254- 3 days post-vaccination | 5 [2.2 to 10.8] | 15 [8.4 to 22.9] | 9 [6.0 to 13.9] | 18 [8.6 to 31.4] | 40 [27.0 to 54.1] | 30 [21.0 to 39.2]
  NZ98/254- 7 days post-vaccination: number analyzed (Participants) | 130 | 103 | 233 | 44 | 54 | 98
  NZ98/254- 7 days post-vaccination | 41 [32.2 to 49.7] | 64 [54.0 to 73.3] | 51 [44.5 to 57.7] | 41 [26.3 to 56.8] | 52 [37.8 to 65.7] | 47 [36.8 to 57.3]
  NZ98/254- 1 month post-vaccination: number analyzed (Participants) | 130 | 103 | 233 | 94 | 109 | 203
  NZ98/254- 1 month post-vaccination | 74 [65.4 to 81.2] | 89 [81.7 to 94.5] | 81 [75.0 to 85.6] | 40 [30.4 to 51.0] | 56 [46.1 to 65.5] | 49 [41.7 to 55.9]
  M10713- 3 days post-vaccination: number analyzed (Participants) | 129 | 112 | 241 | 50 | 55 | 105
  M10713- 3 days post-vaccination | 48 [39.2 to 57.0] | 71 [61.2 to 78.8] | 59 [52.0 to 64.8] | 50 [35.5 to 64.5] | 76 [63.0 to 86.8] | 64 [53.9 to 73.0]
  M10713- 7 days post-vaccination: number analyzed (Participants) | 129 | 112 | 241 | 44 | 54 | 98
  M10713- 7 days post-vaccination | 85 [78.0 to 90.9] | 91 [84.2 to 95.6] | 88 [83.2 to 91.8] | 84 [69.9 to 93.4] | 91 [79.7 to 96.9] | 88 [79.6 to 93.5]
  M10713- 1 month post-vaccination: number analyzed (Participants) | 129 | 112 | 241 | 94 | 109 | 203
  M10713- 1 month post-vaccination | 93 [87.2 to 96.8] | 97 [92.4 to 99.4] | 95 [91.5 to 97.4] | 76 [65.6 to 83.8] | 92 [84.9 to 96.2] | 84 [78.5 to 89.0]
Statistical Analysis 1: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 19, analysis 1]; Test type: Other — Vaccine comparison at Day 4 Group 3B vs Day 34 Group B_0_1 (3 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -30, 95% CI 2-sided [-40.4 to -19.0]
Statistical Analysis 2: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 19, analysis 2]; Test type: Other — Vaccine comparison at Day 8 Group 3B vs Day 38 Group B_0_1 (7 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 3, 95% CI 2-sided [-2.6 to 10.3]
Statistical Analysis 3: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 19, analysis 3]; Test type: Other — Vaccine comparison at Day 31 Group 3B vs Day 61 Group B_0_1 (1 month after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 8, 95% CI 2-sided [3.9 to 12.5]
Statistical Analysis 4: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 19, analysis 1]; Test type: Other — Vaccine comparison at Day 4 Group 3B (V72_41) vs Day 34 Group B_0_1 (V72_41) (3 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -27, 95% CI 2-sided [-41.8 to -12.9]
Statistical Analysis 5: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 19, analysis 2]; Test type: Other — Vaccine comparison at Day 8 Group 3B (V72_41) vs Day 38 Group B_0_1 (V72_41) (7 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 3, 95% CI 2-sided [-6.0 to 16.2]
Statistical Analysis 6: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 19, analysis 3]; Test type: Other — Vaccine comparison at Day 31 Group 3B (V72_41) vs Day 61 Group B_0_1 (V72_41) (1 month after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 7, 95% CI 2-sided [1.4 to 15.2]
Statistical Analysis 7: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 19, analysis 1]; Test type: Other — Vaccine comparison at Day 4 Group 3B (V72P10) vs Day 34 Group B_0_1 (V72P10) (3 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -31, 95% CI 2-sided [-45.1 to -14.6]
Statistical Analysis 8: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 19, analysis 2]; Test type: Other — Vaccine comparison at Day 8 Group 3B (V72P10) vs Day 38 Group B_0_1 (V72P10) (7 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 4, 95% CI 2-sided [1.9 to 13.5]
Statistical Analysis 9: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 19, analysis 3]; Test type: Other — Vaccine comparison at Day 31 Group 3B (V72P10) vs Day 61 Group B_0_1 (V72P10) (1 month after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 8, 95% CI 2-sided [4.4 to 15.0]
Statistical Analysis 10: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 18, analysis 1]; Test type: Other — Vaccine comparison at Day 4 Group 3B vs Day 34 Group B_0_1 (3 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -5, 95% CI 2-sided [-16.0 to 6.5]
Statistical Analysis 11: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 18, analysis 4]; Test type: Other — Vaccine comparison at Day 8 Group 3B vs Day 38 Group B_0_1 (7 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 1, 95% CI 2-sided [-0.9 to 6.2]
Statistical Analysis 12: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 18, analysis 7]; Test type: Other — Vaccine comparison at Day 31 Group 3B vs Day 61 Group B_0_1 (1 month after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 2, 95% CI 2-sided [-0.33 to 5.0]
Statistical Analysis 13: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 18, analysis 1]; Test type: Other — Vaccine comparison at Day 4 Group 3B (V72_41) vs Day 34 Group B_0_1 (V72_41) (3 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -6, 95% CI 2-sided [-20.5 to 10.6]
Statistical Analysis 14: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 18, analysis 4]; Test type: Other — Vaccine comparison at Day 8 Group 3B (V72_41) vs Day 38 Group B_0_1 (V72_41) (7 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 0, 95% CI 2-sided [-3.6 to 8.8]
Statistical Analysis 15: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 18, analysis 7]; Test type: Other — Vaccine comparison at Day 31 Group 3B (V72_41) vs Day 61 Group B_0_1 (V72_41) (1 month after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 0, 95% CI 2-sided [-3.6 to 4.4]
Statistical Analysis 16: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 18, analysis 1]; Test type: Other — Vaccine comparison at Day 4 Group 3B (V72P10) vs Day 34 Group B_0_1 (V72P10) (3 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -4, 95% CI 2-sided [-19.4 to 13.0]
Statistical Analysis 17: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 18, analysis 4]; Test type: Other — Vaccine comparison at Day 8 Group 3B (V72P10) vs Day 38 Group B_0_1 (V72P10) (7 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 2, 95% CI 2-sided [-2.5 to 11.0]
Statistical Analysis 18: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 18, analysis 7]; Test type: Other — Vaccine comparison at Day 31 Group 3B (V72P10) vs Day 61 Group B_0_1 (V72P10) (1 month after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 3, 95% CI 2-sided [-1.2 to 9.4]
Statistical Analysis 19: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 18, analysis 10]; Test type: Other — Vaccine comparison at Day 4 Group 3B vs Day 34 Group B_0_1 (3 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -20, 95% CI 2-sided [-30.0 to -11.1]
Statistical Analysis 20: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 18, analysis 13]; Test type: Other — Vaccine comparison at Day 8 Group 3B vs Day 38 Group B_0_1 (7 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 4, 95% CI 2-sided [-7.6 to 15.7]
Statistical Analysis 21: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 18, analysis 16]; Test type: Other — Vaccine comparison at Day 31 Group 3B vs Day 61 Group B_0_1 (1 month after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 32, 95% CI 2-sided [23.2 to 40.2]
Statistical Analysis 22: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 18, analysis 10]; Test type: Other — Vaccine comparison at Day 4 Group 3B (V72_41) vs Day 34 Group B_0_1 (V72_41) (3 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -13, 95% CI 2-sided [-25.9 to -3.0]
Statistical Analysis 23: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 18, analysis 13]; Test type: Other — Vaccine comparison at Day 8 Group 3B (V72_41) vs Day 38 Group B_0_1 (V72_41) (7 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 0, 95% CI 2-sided [-17.1 to 15.9]
Statistical Analysis 24: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 18, analysis 16]; Test type: Other — Vaccine comparison at Day 31 Group 3B (V72_41) vs Day 61 Group B_0_1 (V72_41) (1 month after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 33, 95% CI 2-sided [20.5 to 45.3]
Statistical Analysis 25: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 18, analysis 10]; Test type: Other — Vaccine comparison at Day 4 Group 3B (V72P10) vs Day 34 Group B_0_1 (V72P10) (3 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -25, 95% CI 2-sided [-40.1 to -11.2]
Statistical Analysis 26: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 18, analysis 13]; Test type: Other — Vaccine comparison at Day 8 Group 3B (V72P10) vs Day 38 Group B_0_1 (V72P10) (7 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 12, 95% CI 2-sided [-3.9 to 28.1]
Statistical Analysis 27: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 18, analysis 16]; Test type: Other — Vaccine comparison at Day 31 Group 3B (V72P10) vs Day 61 Group B_0_1 (V72P10) (1 month after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 33, 95% CI 2-sided [22.0 to 44.1]
Statistical Analysis 28: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 19, analysis 13]; Test type: Other — Vaccine comparison at Day 4 Group 3B vs Day 34 Group B_0_1 (3 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -5, 95% CI 2-sided [-16.0 to 6.0]
Statistical Analysis 29: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 19, analysis 14]; Test type: Other — Vaccine comparison at Day 8 Group 3B vs Day 38 Group B_0_1 (7 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 0, 95% CI 2-sided [-6.8 to 8.9]
Statistical Analysis 30: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 19, analysis 15]; Test type: Other — Vaccine comparison at Day 31 Group 3B vs Day 61 Group B_0_1 (1 month after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 11, 95% CI 2-sided [5.3 to 16.9]
Statistical Analysis 31: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 19, analysis 13]; Test type: Other — Vaccine comparison at Day 4 Group 3B (V72_41) vs Day 34 Group B_0_1 (V72_41) (3 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -2, 95% CI 2-sided [-18.0 to 14.1]
Statistical Analysis 32: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 19, analysis 14]; Test type: Other — Vaccine comparison at Day 8 Group 3B (V72_41) vs Day 38 Group B_0_1 (V72_41) (7 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 1, 95% CI 2-sided [-9.7 to 15.7]
Statistical Analysis 33: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 19, analysis 15]; Test type: Other — Vaccine comparison at Day 31 Group 3B (V72_41) vs Day 61 Group B_0_1 (V72_41) (1 month after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 17, 95% CI 2-sided [8.2 to 27.8]
Statistical Analysis 34: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 19, analysis 13]; Test type: Other — Vaccine comparison at Day 4 Group 3B (V72P10) vs Day 34 Group B_0_1 (V72P10) (3 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = -6, 95% CI 2-sided [-19.1 to 9.1]
Statistical Analysis 35: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 19, analysis 14]; Test type: Other — Vaccine comparison at Day 8 Group 3B (V72P10) vs Day 38 Group B_0_1 (V72P10) (7 days after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 0, 95% CI 2-sided [-8.4 to 11.8]
Statistical Analysis 36: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 19, analysis 15]; Test type: Other — Vaccine comparison at Day 31 Group 3B (V72P10) vs Day 61 Group B_0_1 (V72P10) (1 month after booster or 2nd dose); Miettinen and Nurminen score method; vaccine group difference = 6, 95% CI 2-sided [-0.47 to 12.6]

22. Secondary Outcome: hSBA Geometric Mean Titers Prior to Booster/Second Dose of Vaccination & Post Booster/Second Dose of Vaccination.
Description: as for outcome 20
Time Frame: Group 3B: Day 1 (pre-booster dose) and 3, 7 and 30 days after third dose booster; Group B_0_1: Pre 2nd dose and at 3 (group B_0_1_1 only), 7 (group B_0_1_2 only) and 30 days post second dose.
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 3B (V72_41) | Group 3B (V72P10) | Group 3B | Group B_0_1 (V72_41) | Group B_0_1 (V72P10) | Group B_0_1
Number analyzed (Participants) | 130 | 112 | 242 | 94 | 109 | 203
Titers
  H44/76 - pre-vaccination | 2.41 [1.86 to 3.13] | 4.61 [3.34 to 6.38] | 2.99 [2.41 to 3.70] | 14 [10 to 19] | 27 [19 to 37] | 17 [14 to 22]
  H44/76 - 3 days post-vacc: number analyzed (Participants) | 130 | 112 | 242 | 50 | 55 | 105
  H44/76 - 3 days post-vacc | 2.68 [2.06 to 3.48] | 4.57 [3.38 to 6.18] | 3.20 [2.60 to 3.94] | 14 [9.55 to 22] | 24 [16 to 37] | 17 [13 to 23]
  H44/76 - 7 days post-vacc: number analyzed (Participants) | 130 | 112 | 242 | 44 | 54 | 98
  H44/76 - 7 days post-vacc | 97 [77 to 123] | 153 [123 to 191] | 115 [98 to 136] | 62 [42 to 90] | 60 [44 to 83] | 57 [44 to 73]
  H44/76 - 1 month post-vacc. | 157 [127 to 193] | 285 [234 to 345] | 196 [170 to 228] | 57 [45 to 73] | 64 [52 to 78] | 56 [48 to 66]
  5/99- pre-vaccination: number analyzed (Participants) | 100 | 75 | 175 | 82 | 87 | 169
  5/99- pre-vaccination | 20 [14 to 29] | 30 [20 to 47] | 24 [18 to 32] | 33 [23 to 50] | 30 [20 to 44] | 31 [23 to 41]
  5/99- 3 days post-vacc: number analyzed (Participants) | 103 | 82 | 185 | 44 | 42 | 86
  5/99- 3 days post-vacc | 23 [16 to 34] | 25 [17 to 35] | 24 [18 to 31] | 27 [15 to 49] | 28 [17 to 47] | 27 [19 to 41]
  5/99- 7 days post-vacc: number analyzed (Participants) | 103 | 82 | 185 | 40 | 48 | 88
  5/99- 7 days post-vacc | 1969 [1516 to 2556] | 1547 [1191 to 2009] | 1787 [1477 to 2162] | 294 [197 to 439] | 365 [259 to 514] | 337 [257 to 442]
  5/99- 1 month post-vacc.: number analyzed (Participants) | 103 | 82 | 185 | 84 | 90 | 174
  5/99- 1 month post-vacc. | 2147 [1749 to 2635] | 1903 [1469 to 2466] | 2026 [1714 to 2395] | 224 [179 to 281] | 276 [215 to 353] | 248 [208 to 295]
  NZ98/254- pre-vaccination: number analyzed (Participants) | 130 | 101 | 231 | 93 | 108 | 201
  NZ98/254- pre-vaccination | 1.31 [1.06 to 1.63] | 2.40 [1.72 to 3.37] | 1.57 [1.29 to 1.92] | 3.44 [2.66 to 4.43] | 9.79 [7.07 to 14] | 5.11 [4.10 to 6.38]
  NZ98/254- 3 days post-vacc: number analyzed (Participants) | 130 | 103 | 233 | 50 | 55 | 105
  NZ98/254- 3 days post-vacc | 1.40 [1.15 to 1.70] | 2.34 [1.72 to 3.20] | 1.62 [1.35 to 1.96] | 2.75 [2.02 to 3.74] | 8.94 [5.84 to 14] | 4.45 [3.38 to 5.84]
  NZ98/254- 7 days post-vacc: number analyzed (Participants) | 130 | 103 | 233 | 44 | 54 | 98
  NZ98/254- 7 days post-vacc | 10 [7.80 to 13] | 18 [13 to 25] | 12 [10 to 15] | 11 [6.96 to 17] | 15 [9.79 to 24] | 12 [8.46 to 16]
  NZ98/254- 1 month post-vacc.: number analyzed (Participants) | 130 | 103 | 233 | 94 | 109 | 203
  NZ98/254- 1 month post-vacc. | 32 [25 to 40] | 44 [33 to 59] | 35 [29 to 42] | 12 [9.04 to 16] | 17 [13 to 23] | 14 [11 to 17]
  M10713- pre-vaccination: number analyzed (Participants) | 128 | 112 | 240 | 93 | 109 | 202
  M10713- pre-vaccination | 13 [9.76 to 18] | 22 [16 to 29] | 15 [12 to 19] | 25 [18 to 35] | 50 [38 to 67] | 32 [25 to 41]
  M10713- 3 days post-vacc: number analyzed (Participants) | 129 | 112 | 241 | 50 | 55 | 105
  M10713- 3 days post-vacc | 14 [9.96 to 19] | 24 [18 to 32] | 16 [13 to 21] | 18 [11 to 30] | 37 [24 to 56] | 23 [17 to 33]
  M10713- 7 days post-vacc: number analyzed (Participants) | 129 | 112 | 241 | 44 | 54 | 98
  M10713- 7 days post-vacc | 48 [39 to 59] | 68 [56 to 82] | 54 [46 to 62] | 42 [30 to 59] | 56 [42 to 73] | 45 [36 to 57]
  M10713- 1 month post-vacc.: number analyzed (Participants) | 129 | 112 | 241 | 94 | 109 | 203
  M10713- 1 month post-vacc. | 64 [52 to 80] | 116 [94 to 143] | 78 [67 to 92] | 34 [26 to 44] | 61 [49 to 75] | 41 [35 to 49]
Statistical Analysis 1: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 6, analysis 1]; Test type: Other — Vaccine Comparison Day 31 Group 3B vs Day 61 Group B_0_1(1 month after booster or 2nd dose); ANOVA; Ratio of GMTs = 3.49, 95% CI 2-sided [2.85 to 4.29]
Statistical Analysis 2: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 6, analysis 1]; Test type: Other — Vaccine Comparison Day 31 Group 3B (V72_41) vs Day 61 Group B_0_1 (V72_41) (1 month after booster or 2nd dose); ANOVA; Ratio of GMTs = 2.73, 95% CI 2-sided [2.02 to 3.69]
Statistical Analysis 3: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 6, analysis 1]; Test type: Other — Vaccine Comparison Day 31 Group 3B (V72P10) vs Day 61 Group B_0_1 (V72P10) (1 month after booster or 2nd dose); ANOVA; Ratio of GMTs = 4.46, 95% CI 2-sided [3.38 to 5.88]
Statistical Analysis 4: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 6, analysis 4]; Test type: Other — Vaccine Comparison Day 31 Group 3B vs Day 61 Group B_0_1(1 month after booster or 2nd dose); ANOVA; Ratio of GMTs = 8.18, 95% CI 2-sided [6.51 to 10]
Statistical Analysis 5: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 6, analysis 4]; Test type: Other — Vaccine Comparison Day 31 Group 3B (V72_41) vs Day 61 Group B_0_1 (V72_41) (1 month after booster or 2nd dose); ANOVA; Ratio of GMTs = 9.58, 95% CI 2-sided [7.17 to 13]
Statistical Analysis 6: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 6, analysis 4]; Test type: Other — Vaccine Comparison Day 31 Group 3B (V72P10) vs Day 61 Group B_0_1 (V72P10) (1 month after booster or 2nd dose); ANOVA; Ratio of GMTs = 6.90, 95% CI 2-sided [4.82 to 9.87]
Statistical Analysis 7: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 6, analysis 7]; Test type: Other — Vaccine Comparison Day 31 Group 3B vs Day 61 Group B_0_1(1 month after booster or 2nd dose); ANOVA; Ratio of GMTs = 2.58, 95% CI 2-sided [1.98 to 3.36]
Statistical Analysis 8: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 6, analysis 7]; Test type: Other — Vaccine Comparison Day 31 Group 3B (V72_41) vs Day 61 Group B_0_1 (V72_41) (1 month after booster or 2nd dose); ANOVA; Ratio of GMTs = 2.65, 95% CI 2-sided [1.89 to 3.73]
Statistical Analysis 9: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 6, analysis 7]; Test type: Other — Vaccine Comparison Day 31 Group 3B (V72P10) vs Day 61 Group B_0_1 (V72P10) (1 month after booster or 2nd dose); ANOVA; Ratio of GMTs = 2.51, 95% CI 2-sided [1.67 to 3.78]
Statistical Analysis 10: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 6, analysis 10]; Test type: Other — Vaccine Comparison Day 31 Group 3B vs Day 61 Group B_0_1(1 month after booster or 2nd dose); ANOVA; Ratio of GMTs = 1.90, 95% CI 2-sided [1.52 to 2.36]
Statistical Analysis 11: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 6, analysis 10]; Test type: Other — Vaccine Comparison Day 31 Group 3B (V72_41) vs Day 61 Group B_0_1 (V72_41) (1 month after booster or 2nd dose); ANOVA; Ratio of GMTs = 1.88, 95% CI 2-sided [1.37 to 2.59]
Statistical Analysis 12: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 6, analysis 10]; Test type: Other — Vaccine Comparison Day 31 Group 3B (V72P10) vs Day 61 Group B_0_1 (V72P10) (1 month after booster or 2nd dose); ANOVA; Ratio of GMTs = 1.91, 95% CI 2-sided [1.41 to 2.58]

23. Secondary Outcome: Geometric Mean Ratios (GMRs) of GMTs After Booster/Second Vaccination Versus Before Booster/Second Vaccination.
Description: Bactericidal activity was measured against each of the four N. meningitidis group B indicator strains H44/76,5/99,NZ98/254 and M10713 by calculating the GMRs of GMTs post-vaccination with a booster dose (Group 3B) versus pre-booster dose or second dose (Group B_0_1) of vaccination versus pre second dose.
Time Frame: Group 3B: Day 1 and 30 days after third dose booster; Group B_0_1: 30 days post-first dose and at 30 days post-second dose
Population: as for outcome 20
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Group 3B (V72_41) | Group 3B (V72P10) | Group 3B | Group B_0_1 (V72_41) | Group B_0_1 (V72P10) | Group B_0_1
Number analyzed (Participants) | 130 | 112 | 242 | 94 | 109 | 203
Ratio
  H44/76 | 65 [49 to 85] | 62 [49 to 78] | 66 [55 to 79] | 4.21 [3.05 to 5.80] | 2.37 [1.87 to 3.00] | 3.27 [2.66 to 4.03]
  5/99: number analyzed (Participants) | 100 | 75 | 175 | 82 | 87 | 169
  5/99 | 105 [76 to 145] | 62 [41 to 96] | 85 [65 to 111] | 6.86 [4.82 to 9.78] | 9.09 [6.10 to 14] | 8.10 [6.12 to 11]
  NZ98/25: number analyzed (Participants) | 130 | 101 | 231 | 93 | 108 | 201
  NZ98/25 | 24 [19 to 30] | 18 [14 to 24] | 22 [19 to 27] | 3.42 [2.59 to 4.51] | 1.76 [1.36 to 2.29] | 2.63 [2.15 to 3.21]
  M10713: number analyzed (Participants) | 128 | 112 | 240 | 93 | 109 | 202
  M10713 | 4.87 [3.92 to 6.05] | 5.30 [4.29 to 6.55] | 5.07 [4.33 to 5.94] | 1.36 [1.06 to 1.75] | 1.20 [0.97 to 1.49] | 1.27 [1.07 to 1.52]

24. Secondary Outcome: Percentages of Subjects With at Least Four-fold Increase in hSBA Titers Pre-booster/Second Dose Vaccination- Compared to 3, 7 and 30 Days Post- Booster/Second Vaccination
Description: The percentage of subjects with 4-fold rise at 3, 7, 30 days post-vaccination with a booster dose (follow-on subjects) /second dose (naive subjects) of rMenB+OMV NZ with respect to day 1 (follow-on subjects) / pre-second dose of rMenB+OMV NZ (naïve subjects). Percentage of subjects with four-fold rise in hSBA titers relative to baseline were defined as: • for a pre-vaccination titer < 4, a post-vaccination titer of at least 16; • for a pre-vaccination titer ≥ 4 but <LLOQ, a post vaccination titer of at least fourfold the LLOQ; • for a pre-vaccination titer ≥LLOQ, a post vaccination titer of at least fourfold the pre-vaccination titer.
Time Frame: Group 3B: at 3, 7 and 30 days after third dose booster; Group B_0_1: at 3 (group B_0_1_1 only), 7 (group B_0_1_2 only) and 30 days post second dose
Population: Analysis was performed on PPS kinetics which included all subjects who had no protocol deviations/any other reason defined prior to analysis, leading to exclusion & correctly received the vaccination at day 1/day 31 & day 1 & provided evaluable immunogenicity result at all of days 4, 8 & 31 (follow-on subjects)or at all of days 34/38 & 61(naive)
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Group 3B (V72_41) | Group 3B (V72P10) | Group 3B | Group B_0_1 (V72_41) | Group B_0_1 (V72P10) | Group B_0_1
Number analyzed (Participants) | 130 | 112 | 242 | 94 | 109 | 203
Percentage of subjects
  H44/76 3 days post vaccination: number analyzed (Participants) | 130 | 112 | 242 | 50 | 55 | 105
  H44/76 3 days post vaccination | 2 [0.48 to 6.6] | 2 [0.22 to 6.3] | 2 [0.7 to 4.8] | 6 [1.3 to 16.5] | 2 [0.05 to 9.7] | 4 [1.0 to 9.5]
  H44/76 - 7 days post-vacc: number analyzed (Participants) | 130 | 112 | 242 | 44 | 54 | 98
  H44/76 - 7 days post-vacc | 89 [82.6 to 94.0] | 86 [77.8 to 91.6] | 88 [82.8 to 91.5] | 45 [30.4 to 61.2] | 26 [15.0 to 39.7] | 35 [25.4 to 45.0]
  H44/76 - 1 month post-vacc. | 95 [89.2 to 97.8] | 98 [93.7 to 99.78] | 96 [93.1 to 98.3] | 51 [40.5 to 61.5] | 28 [19.4 to 36.9] | 38 [31.7 to 45.5]
  5/99- 3 days post-vacc: number analyzed (Participants) | 100 | 75 | 175 | 44 | 39 | 83
  5/99- 3 days post-vacc | 7 [2.9 to 13.9] | 1 [0.03 to 7.2] | 5 [2.0 to 8.8] | 5 [0.6 to 15.5] | 8 [1.6 to 20.9] | 6 [2.0 to 13.5]
  5/99- 7 days post-vacc: number analyzed (Participants) | 100 | 75 | 175 | 38 | 48 | 86
  5/99- 7 days post-vacc | 98 [93.0 to 99.76] | 95 [86.9 to 98.5] | 97 [92.7 to 98.7] | 55 [38.3 to 71.4] | 63 [47.4 to 76.0] | 59 [48.2 to 69.8]
  5/99- 1 month post-vacc.: number analyzed (Participants) | 100 | 75 | 175 | 82 | 87 | 169
  5/99- 1 month post-vacc. | 98 [93.0 to 99.76] | 96 [88.8 to 99.2] | 97 [93.5 to 99.1] | 56 [44.7 to 67.0] | 72 [61.8 to 81.5] | 64 [56.8 to 71.7]
  NZ98/254- 3 days post-vacc: number analyzed (Participants) | 130 | 101 | 231 | 50 | 54 | 104
  NZ98/254- 3 days post-vacc | 2 [0.48 to 6.6] | 2 [0.24 to 7.0] | 2 [0.7 to 5.0] | 2 [0.05 to 10.6] | 2 [0.05 to 9.9] | 2 [0.23 to 6.8]
  NZ98/254- 7 days post-vacc: number analyzed (Participants) | 130 | 101 | 231 | 43 | 54 | 97
  NZ98/254- 7 days post-vacc | 55 [45.7 to 63.4] | 55 [45.2 to 65.3] | 55 [48.3 to 61.5] | 26 [13.5 to 41.2] | 13 [5.4 to 24.9] | 19 [11.4 to 27.7]
  NZ98/254- 1 month post-vacc.: number analyzed (Participants) | 130 | 101 | 231 | 93 | 108 | 201
  NZ98/254- 1 month post-vacc. | 82 [73.8 to 87.8] | 80 [71.1 to 87.5] | 81 [75.3 to 85.8] | 35 [25.8 to 46.1] | 20 [13.2 to 29.2] | 27 [21.3 to 34.1]
  M10713- 3 days post-vacc: number analyzed (Participants) | 128 | 112 | 240 | 50 | 55 | 105
  M10713- 3 days post-vacc | 2 [0.49 to 6.7] | 3 [0.6 to 7.6] | 3 [0.9 to 5.4] | 0 [0.0 to 7.1] | 0 [0.0 to 6.5] | 0 [0.0 to 3.5]
  M10713- 7 days post-vacc: number analyzed (Participants) | 128 | 112 | 240 | 43 | 54 | 97
  M10713- 7 days post-vacc | 39 [30.6 to 48.1] | 28 [19.6 to 36.9] | 34 [27.8 to 40.1] | 14 [5.3 to 27.9] | 0 [0.0 to 6.6] | 6 [2.3 to 13.0]
  M10713- 1 month post-vacc.: number analyzed (Participants) | 128 | 112 | 240 | 93 | 109 | 202
  M10713- 1 month post-vacc. | 48 [39.5 to 57.4] | 49 [39.5 to 58.7] | 49 [42.3 to 55.3] | 12 [6.1 to 20.2] | 7 [3.2 to 14.0] | 9 [5.8 to 14.3]
Statistical Analysis 1: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 19, analysis 1]; Test type: Other — 3 Days Post Booster/Second Vaccination. Four-fold Increase (Group 3B vs. Group B_0_1) Difference; Miettinen and Nurminen score method; Vaccine group difference = -2, 95% CI 2-sided [-7.5 to 1.8]
Statistical Analysis 2: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 19, analysis 2]; Test type: Other — 7 Days Post Booster/Second Vaccination. Four-fold Increase (Group 3B vs. Group B_0_1) Difference; Miettinen and Nurminen score method; vaccine group difference = 53, 95% CI 2-sided [42.1 to 62.5]
Statistical Analysis 3: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 19, analysis 3]; Test type: Other — 1 Month Post Booster/Second Vaccination. Four-fold Increase (Group 3B vs. Group B_0_1) Difference; Miettinen and Nurminen score method; vaccine group difference = 58, 95% CI 2-sided [50.5 to 64.7]
Statistical Analysis 4: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 19, analysis 1]; Test type: Other — 3 Days Post Booster/Second Vaccination. Four-fold Increase [Group 3B (V72_41) vs. Group B_0_1 (V72_41)] Difference; Miettinen and Nurminen score method; vaccine group difference = -4, 95% CI 2-sided [-14.1 to 2.0]
Statistical Analysis 5: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 19, analysis 2]; Test type: Other — 7 Days Post Booster/Second Vaccination. Four-fold Increase [Group 3B (V72_41) vs. Group B_0_1 (V72_41)] Difference; Miettinen and Nurminen score method; vaccine group difference = 44, 95% CI 2-sided [28.1 to 58.5]
Statistical Analysis 6: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 19, analysis 3]; Test type: Other — 1 month Post Booster/Second Vaccination. Four-fold Increase [Group 3B (V72_41) vs. Group B_0_1 (V72_41)] Difference; Miettinen and Nurminen score method; vaccine group difference = 44, 95% CI 2-sided [32.7 to 54.1]
Statistical Analysis 7: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 19, analysis 1]; Test type: Other — 3 Days Post Booster/Second Vaccination. Four-fold Increase [Group 3B (V72P10) vs. Group B_0_1 (V72P10)] Difference; Miettinen and Nurminen score method; vaccine group difference = 0, 95% CI 2-sided [-8.0 to 4.8]
Statistical Analysis 8: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 19, analysis 2]; Test type: Other — 7 Days Post Booster/Second Vaccination. Four-fold Increase [Group 3B (V72P10) vs. Group B_0_1 (V72P10)] Difference; Miettinen and Nurminen score method; Vaccine group difference = 60, 95% CI 2-sided [45.0 to 71.5]
Statistical Analysis 9: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 19, analysis 3]; Test type: Other — 1 month Post Booster/Second Vaccination. Four-fold Increase [Group 3B (V72P10) vs. Group B_0_1 (V72P10)] Difference; Miettinen and Nurminen score method; vaccine group difference = 71, 95% CI 2-sided [61.2 to 78.5]
Statistical Analysis 10: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 18, analysis 1]; Test type: Other — 3 Days Post Booster/Second Vaccination. Four-fold Increase (Group 3B vs. Group B_0_1) Difference; Miettinen and Nurminen score method; vaccine group difference = -1, 95% CI 2-sided [-9.1 to 4]
Statistical Analysis 11: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 18, analysis 4]; Test type: Other — 7 Days Post Booster/Second Vaccination. Four-fold Increase (Group 3B vs. Group B_0_1) Difference; Miettinen and Nurminen score method; vaccine group difference = 37, 95% CI 2-sided [27.0 to 48.1]
Statistical Analysis 12: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 18, analysis 7]; Test type: Other — 1 Month Post Booster/Second Vaccination. Four-fold Increase (Group 3B vs. Group B_0_1) Difference; Miettinen and Nurminen score method; Vaccine group difference = 33, 95% CI 2-sided [25.2 to 40.4]
Statistical Analysis 13: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 18, analysis 1]; Test type: Other — 3 Days Post Booster/Second Vaccination. Four-fold Increase [Group 3B (V72_41) vs. Group B_0_1 (V72_41)] Difference; Miettinen and Nurminen score method; vaccine group difference = 2, 95% CI 2-sided [-8.7 to 10.2]
Statistical Analysis 14: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 18, analysis 4]; Test type: Other — 7 Days Post Booster/Second Vaccination. Four-fold Increase [Group 3B (V72_41) vs. Group B_0_1 (V72_41)] Difference; Miettinen and Nurminen score method; vaccine group difference = 43, 95% CI 2-sided [27.7 to 58.6]
Statistical Analysis 15: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 18, analysis 7]; Test type: Other — 1 month Post Booster/Second Vaccination. Four-fold Increase [Group 3B (V72_41) vs. Group B_0_1 (V72_41)] Difference; Miettinen and Nurminen score method; vaccine group difference = 42, 95% CI 2-sided [31.1 to 53.0]
Statistical Analysis 16: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 18, analysis 1]; Test type: Other — 3 Days Post Booster/Second Vaccination. Four-fold Increase [Group 3B (V72P10) vs. Group B_0_1 (V72P10)] Difference; Miettinen and Nurminen score method; vaccine group difference = -6, 95% CI 2-sided [-19.2 to 0.9]
Statistical Analysis 17: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 18, analysis 4]; Test type: Other — 7 Days Post Booster/Second Vaccination. Four-fold Increase [Group 3B (V72P10) vs. Group B_0_1 (V72P10)] Difference; Miettinen and Nurminen score method; vaccine group difference = 32, 95% CI 2-sided [18.2 to 47.0]
Statistical Analysis 18: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 18, analysis 7]; Test type: Other — 1 month Post Booster/Second Vaccination. Four-fold Increase [Group 3B (V72P10) vs. Group B_0_1 (V72P10)] Difference; Miettinen and Nurminen score method; vaccine group difference = 24, 95% CI 2-sided [13.2 to 34.4]
Statistical Analysis 19: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 18, analysis 10]; Test type: Other — 3 Days Post Booster/Second Vaccination. Four-fold Increase (Group 3B vs. Group B_0_1) Difference; Miettinen and Nurminen score method; vaccine group difference = 0, 95% CI 2-sided [-4.7 to 3.4]
Statistical Analysis 20: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 18, analysis 13]; Test type: Other — 7 Days Post Booster/Second Vaccination. Four-fold Increase (Group 3B vs. Group B_0_1) Difference; Miettinen and Nurminen score method; Vaccine group difference = 36, 95% CI 2-sided [25.6 to 45.7]
Statistical Analysis 21: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 18, analysis 16]; Test type: Other — 1 Month Post Booster/Second Vaccination. Four-fold Increase (Group 3B vs. Group B_0_1) Difference; Miettinen and Nurminen score method; vaccine group difference = 54, 95% CI 2-sided [45.2 to 61.1]
Statistical Analysis 22: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 18, analysis 10]; Test type: Other — 3 Days Post Booster/Second Vaccination. Four-fold Increase [Group 3B (V72_41) vs. Group B_0_1 (V72_41)] Difference; Miettinen and Nurminen score method; vaccine group difference = 0, 95% CI 2-sided [-8.4 to 5.0]
Statistical Analysis 23: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 18, analysis 13]; Test type: Other — 7 Days Post Booster/Second Vaccination. Four-fold Increase [Group 3B (V72_41) vs. Group B_0_1 (V72_41)] Difference; Miettinen and Nurminen score method; vaccine group difference = 29, 95% CI 2-sided [12.1 to 43.0]
Statistical Analysis 24: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); 1 month post vaccination-The group difference in percentages of subjects with response against N. meningitidis serogroup B indicator strain NZ98/154 and the associated confidence interval for the difference was calculated using the method of Miettinen and Nurminen; Test type: Other — 1 month Post Booster/Second Vaccination. Four-fold Increase [Group 3B (V72_41) vs. Group B_0_1 (V72_41)] Difference; Miettinen and Nurminen score method; Vaccine group difference = 46, 95% CI 2-sided [33.6 to 57.1]
Statistical Analysis 25: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 18, analysis 10]; Test type: Other — 3 Days Post Booster/Second Vaccination. Four-fold Increase [Group 3B (V72P10) vs. Group B_0_1 (V72P10)] Difference; Miettinen and Nurminen score method; Vaccine group difference = 0, 95% CI 2-sided [-8.0 to 5.4]
Statistical Analysis 26: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 18, analysis 13]; Test type: Other — 7 Days Post Booster/Second Vaccination. Four-fold Increase [Group 3B (V72P10) vs. Group B_0_1 (V72P10)] Difference; Miettinen and Nurminen score method; Vaccine group difference = 42, 95% CI 2-sided [27.8 to 54.5]
Statistical Analysis 27: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 18, analysis 16]; Test type: Other — 1 month Post Booster/Second Vaccination. Four-fold Increase [Group 3B (V72P10) vs. Group B_0_1 (V72P10)] Difference; Miettinen and Nurminen score method; vaccine group difference = 60, 95% CI 2-sided [47.9 to 69.6]
Statistical Analysis 28: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 19, analysis 13]; Test type: Other — 3 Days Post Booster/Second Vaccination. Four-fold Increase (Group 3B vs. Group B_0_1) Difference; Miettinen and Nurminen score method; vaccine group difference = 3, 95% CI 2-sided [-1.1 to 5.4]
Statistical Analysis 29: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 19, analysis 14]; Test type: Other — 7 Days Post Booster/Second Vaccination. Four-fold Increase (Group 3B vs. Group B_0_1) Difference; Miettinen and Nurminen score method; vaccine group difference = 28, 95% CI 2-sided [19.1 to 34.9]
Statistical Analysis 30: Comparison: Group 3B vs Group B_0_1; [analysis description as in outcome 19, analysis 15]; Test type: Other — 1 Month Post Booster/Second Vaccination. Four-fold Increase (Group 3B vs. Group B_0_1) Difference; Miettinen and Nurminen score method; vaccine group difference = 39, 95% CI 2-sided [31.6 to 46.6]
Statistical Analysis 31: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 19, analysis 13]; Test type: Other — 3 Days Post Booster/Second Vaccination. Four-fold Increase [Group 3B (V72_41) vs. Group B_0_1 (V72_41)] Difference; Miettinen and Nurminen score method; Vaccine group difference = 2, 95% CI 2-sided [-4.9 to 6.7]
Statistical Analysis 32: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 19, analysis 14]; Test type: Other — 7 Days Post Booster/Second Vaccination. Four-fold Increase [Group 3B (V72_41) vs. Group B_0_1 (V72_41)] Difference; Miettinen and Nurminen score method; Vaccine group difference = 25, 95% CI 2-sided [9.7 to 37.1]
Statistical Analysis 33: Comparison: Group 3B (V72_41) vs Group B_0_1 (V72_41); [analysis description as in outcome 19, analysis 15]; Test type: Other — 1 month Post Booster/Second Vaccination. Four-fold Increase [Group 3B (V72_41) vs. Group B_0_1 (V72_41)] Difference; Miettinen and Nurminen score method; Vaccine group difference = 37, 95% CI 2-sided [25.1 to 47.0]
Statistical Analysis 34: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 19, analysis 13]; Test type: Other — 3 Days Post Booster/Second Vaccination. Four-fold Increase [Group 3B (V72P10) vs. Group B_0_1 (V72P10)] Difference; Miettinen and Nurminen score method; Vaccine group difference = 3, 95% CI 2-sided [-3.9 to 7.6]
Statistical Analysis 35: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 19, analysis 14]; Test type: Other — 7 Days Post Booster/Second Vaccination. Four-fold Increase [Group 3B (V72P10) vs. Group B_0_1 (V72P10)] Difference; Miettinen and Nurminen score method; Vaccine group difference = 28, 95% CI 2-sided [20.2 to 36.6]
Statistical Analysis 36: Comparison: Group 3B (V72P10) vs Group B_0_1 (V72P10); [analysis description as in outcome 19, analysis 15]; Test type: Other — 1 month Post Booster/Second Vaccination. Four-fold Increase [Group 3B (V72P10) vs. Group B_0_1 (V72P10)] Difference; Miettinen and Nurminen score method; Vaccine group difference = 42, 95% CI 2-sided [31.0 to 51.9]

25. Secondary Outcome: Percentage of Subjects With hSBA ≥1:4 After Second Vaccination of rMenB+OMV NZ
Description: Bactericidal activity was measured against the N. meningitidis group B indicator strains 5/99 and NZ98/254. Only subjects receiving a second vaccination (group B_0_1) were assessed for this outcome measure.
Time Frame: At Day 61 (30 days post second dose of vaccination.)
Population: Analysis was performed on the PPS( per protocol set) catch up. The PPS catch up included all subjects who were randomized to group B_0_1 who correctly received two vaccinations at day 1 and day 31 & provided evaluable immunogenicity result at day 61 for atleast one indicator strain. The analysis was performed only on strains 5/99 and NZ98/254
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Group B_0_1 (V72_41) | Group B_0_1 (V72P10) | Group B_0_1
Number analyzed (Participants) | 98 | 117 | 215
Percentage of subjects
  5/99: number analyzed (Participants) | 91 | 104 | 195
  5/99 | 100 [96.0 to 100.0] | 97 [91.8 to 99.4] | 98 [95.6 to 99.68]
  NZ98/254 | 82 [72.5 to 88.7] | 79 [71.0 to 86.4] | 80 [74.5 to 85.5]

26. Secondary Outcome: Percentage of Subjects With hSBA ≥1:5 After Second Vaccination of rMenB+OMV NZ
Description: Bactericidal activity was measured against each of the four N. meningitidis group B indicator strains H44/76 and M10713. Only subjects receiving a second vaccination (group B_0_1) were assessed for this outcome measure.
Time Frame: At Day 61 (30 days post second dose of vaccination.)
Population: Analysis was performed on the PPS( per protocol set) catch up. The PPS catch up included all subjects who were randomized to group B_0_1 who correctly received two vaccinations at day 1 and day 31 & provided evaluable immunogenicity result at day 61 for atleast one indicator strain. The analysis was performed only on strains H44/76 and M10713
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Group B_0_1 (V72_41) | Group B_0_1 (V72P10) | Group B_0_1
Number analyzed (Participants) | 98 | 117 | 215
Percentage of subjects
  H44/76 | 99 [94.4 to 99.97] | 99 [95.3 to 99.98] | 99 [96.7 to 99.89]
  M10713: number analyzed (Participants) | 98 | 116 | 214
  M10713 | 90 [82.0 to 95.0] | 96 [90.2 to 98.6] | 93 [88.7 to 96.0]

27. Secondary Outcome: Percentage of Subjects With hSBA ≥1:8 After Second Vaccination of rMenB+OMV NZ.
Description: Bactericidal activity was measured against each of the four N. meningitidis group B indicator strains H44/76,5/99,NZ98/254 and M10713.
  Only subjects receiving a second vaccination (group B_0_1) were assessed for this outcome measure.
Time Frame: At Day 61 (30 days post second vaccination)
Population: Analysis was performed on the PPS( per protocol set) catch up. The PPS catch up included all subjects who were randomized to group B_0_1 who correctly received two vaccinations at day 1 and day 31 & provided evaluable immunogenicity result at day 61 for atleast one indicator strain.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Group B_0_1 (V72_41) | Group B_0_1 (V72P10) | Group B_0_1
Number analyzed (Participants) | 98 | 117 | 215
Percentage of subjects
  H44/76 | 99 [94.4 to 99.97] | 97 [92.7 to 99.5] | 98 [95.3 to 99.5]
  5/99: number analyzed (Participants) | 91 | 104 | 195
  5/99 | 100 [96.0 to 100.0] | 97 [91.8 to 99.4] | 98 [95.6 to 99.68]
  NZ98/254 | 64 [54.0 to 73.7] | 69 [60.0 to 77.4] | 67 [60.3 to 73.2]
  M10713: number analyzed (Participants) | 98 | 116 | 214
  M10713 | 86 [77.2 to 92.0] | 94 [88.0 to 97.5] | 90 [85.4 to 93.8]

28. Secondary Outcome: Percentage of Subjects With hSBA ≥1:16 After Second Vaccination of rMenB+OMV NZ.
Description: as for outcome 27
Time Frame: At Day 61 (30 days post second vaccination)
Population: as for outcome 27
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Group B_0_1 (V72_41) | Group B_0_1 (V72P10) | Group B_0_1
Number analyzed (Participants) | 98 | 117 | 215
Percentage of subjects
  H44/76 | 91 [83.3 to 95.7] | 91 [83.8 to 95.2] | 91 [86.0 to 94.2]
  5/99: number analyzed (Participants) | 91 | 104 | 195
  5/99 | 100 [96.0 to 100] | 96 [90.4 to 98.9] | 98 [94.8 to 99.4]
  NZ98/254 | 40 [30.0 to 50.2] | 56 [46.1 to 64.7] | 48 [41.5 to 55.3]
  M10713: number analyzed (Participants) | 98 | 116 | 214
  M10713 | 74 [64.7 to 82.8] | 92 [85.8 to 96.4] | 84 [78.5 to 88.7]

29. Secondary Outcome: hSBA Geometric Mean Titers (GMTs) After Second Vaccination of rMenB+OMV NZ.
Description: as for outcome 27
Time Frame: At Day 1 & Day 61 (30 days post second dose of vaccination)
Population: as for outcome 27
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group B_0_1 (V72_41) | Group B_0_1 (V72P10) | Group B_0_1
Number analyzed (Participants) | 98 | 117 | 215
Titers
  H44/76 Day 1 | 1.08 [1.00 to 1.17] | 1.56 [1.29 to 1.89] | 1.32 [1.18 to 1.47]
  H44/76 1 month post 2nd vaccination | 57 [47 to 68] | 64 [53 to 78] | 61 [53 to 70]
  5/99 Day 1: number analyzed (Participants) | 86 | 95 | 181
  5/99 Day 1 | 1.18 [1.03 to 1.35] | 2.18 [1.58 to 3.00] | 1.63 [1.35 to 1.96]
  5/99 1 month post 2nd vaccination: number analyzed (Participants) | 91 | 104 | 195
  5/99 1 month post 2nd vaccination | 239 [200 to 285] | 274 [207 to 363] | 257 [217 to 305]
  NZ98/254 Day 1: number analyzed (Participants) | 98 | 115 | 213
  NZ98/254 Day 1 | 1.00 [1.00 to 1.00] | 1.58 [1.30 to 1.91] | 1.28 [1.15 to 1.42]
  NZ98/254 1 month post 2nd vaccination | 11 [8.41 to 14] | 18 [13 to 24] | 14 [11 to 17]
  M10713 Day 1: number analyzed (Participants) | 98 | 116 | 214
  M10713 Day 1 | 10 [7.13 to 15] | 19 [14 to 26] | 14 [11 to 18]
  M10713 1 month post 2nd vaccination: number analyzed (Participants) | 98 | 116 | 214
  M10713 1 month post 2nd vaccination | 33 [25 to 44] | 60 [48 to 75] | 46 [38 to 55]

30. Secondary Outcome: Geometric Mean Ratio (GMRs) of GMTs One Month Post Second Vaccination Versus Pre Vaccination at Day 1
Description: as for outcome 27
Time Frame: At Day 1 & Day 61 (30 days post 2nd vaccination)
Population: as for outcome 27
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Group B_0_1 (V72_41) | Group B_0_1 (V72P10) | Group B_0_1
Number analyzed (Participants) | 98 | 117 | 215
Ratio
  H44/76 | 52 [42 to 65] | 41 [33 to 51] | 46 [39 to 54]
  5/99: number analyzed (Participants) | 86 | 95 | 181
  5/99 | 204 [162 to 257] | 123 [74 to 204] | 156 [117 to 209]
  NZ98/254: number analyzed (Participants) | 98 | 115 | 213
  NZ98/254 | 11 [8.41 to 14] | 11 [7.94 to 16] | 11 [8.88 to 14]
  M10713: number analyzed (Participants) | 98 | 116 | 214
  M10713 | 3.24 [2.57 to 4.08] | 3.22 [2.60 to 3.98] | 3.23 [2.76 to 3.77]

31. Secondary Outcome: Percentages of Subjects With at Least Four-fold Increase in hSBA Titers at Pre-First Vaccination Compared to One Month Post-Second Vaccination
Description: The percentage of subjects with 4-fold rise at one month post-vaccination with a second dose (naïve subjects) of rMenB+OMV NZ with respect to day 1, to each and any one, two, three or all 4 indicator strains.
  Percentage of subjects with four-fold rise in hSBA titers relative to baseline were defined as:
  * for a pre-vaccination titer < 4, a post-vaccination titer of at least 16;
  * for a pre-vaccination titer ≥ 4 but <LLOQ, a post vaccination titer of at least fourfold the LLOQ;
  * for a pre-vaccination titer ≥LLOQ, a post vaccination titer of at least fourfold the pre-vaccination titer.
  Only subjects receiving the second dose of vaccination(group B_0_1) were considered for this outcome measure.
Time Frame: At Day 61 (30 days post second dose of vaccination)
Population: as for outcome 27
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | Group B_0_1 (V72_41) | Group B_0_1 (V72P10) | Group B_0_1
Number analyzed (Participants) | 98 | 117 | 215
Percentage of Subjects
  H44/76 | 97 [91.3 to 99.4] | 94 [88.1 to 97.6] | 95 [91.6 to 97.7]
  5/99: number analyzed (Participants) | 86 | 95 | 181
  5/99 | 100 [95.8 to 100] | 94 [86.8 to 97.6] | 97 [92.9 to 98.8]
  NZ98/254: number analyzed (Participants) | 98 | 115 | 213
  NZ98/254 | 64 [54.0 to 73.7] | 69 [59.4 to 77.0] | 67 [59.9 to 73]
  M10713: number analyzed (Participants) | 98 | 116 | 214
  M10713 | 37 [27.2 to 47.1] | 33 [24.3 to 42.1] | 35 [28.2 to 41.4]

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected until 7 days after vaccinations. Unsolicited AEs were collected 30 days after each vaccination at day 31 (all subjects) and at day 61 (group B_0_1 subjects only).
Description: Serious Adverse Events (SAEs) were collected until study termination (1 month for group 3B subjects/ 2 months for group B_0_1 subjects)
Groups:
- Group 3B: Subjects who received two doses of rMenB+OMV NZ administered at 0, 1 month schedule in studies V72_41 or V72P10, and who received a third dose booster of rMenB+OMV NZ at 4 to 7.5 years after the last dose received during parent studies, and had blood collected at baseline and at 3, 7 and 30 days after the third dose booster.
- Group B_0_1: Naive subjects from V72_41 or V72P10 studies, who received two doses of rMenB+OMV NZ at a 0 and 1 month schedule and had blood collected at baseline, 30 days after the first dose and 3 or 7, and 30 days after the second dose.
Arm/Group | Group 3B | Group B_0_1
All-Cause Mortality (participants affected / at risk) | 0/275 | 0/255
Serious Adverse Events (participants affected / at risk) | 0/275 | 1/255
Other Adverse Events (participants affected / at risk) | 266/275 | 253/255
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 3B (N=275) | Group B_0_1 (N=255)
Appendicitis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 3B (N=275) | Group B_0_1 (N=255)
Nausea (Gastrointestinal disorders) | 56 | 53
Injectioon site pain (General disorders) | 259 | 251
Injection site erythema (General disorders) | 162 | 135
Fatigue (General disorders) | 156 | 141
Injection site induration (General disorders) | 135 | 136
Injection site swelling (General disorders) | 123 | 111
Pyrexia (General disorders) | 17 | 9
Viral upper respiratory tract infection (Infections and infestations) | 13 | 23
Myalgia (Musculoskeletal and connective tissue disorders) | 121 | 100
Arthralgia (Musculoskeletal and connective tissue disorders) | 85 | 63
Headache (Nervous system disorders) | 150 | 126

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.